

# AtriCure, Inc. 7555 Innovation Way Mason, Ohio 45040

# Long-Term Follow-Up On LAA Exclusion Using AtriClip VCLIP POST-MARKET STUDY CLINICAL TRIAL PROTOCOL: CP-2021-03

| Revision Number | В |
|---|---|
| Date | October 15, 2021 |
| National Principal<br>Investigator/Lead Principal<br>Investigator: | Elias Zias, MD NYU Langone Health 530 1st Ave, NY, NY 10016 Elias.Zias@nyulangone.org |
| Study Oversight Committee | National PI(s) & AtriCure Medical Advisor |
| Planned Number of Sites and Region(s) (US/OUS) | Up to 170 subjects will be enrolled at up to 20 sites in the US, United Kingdom (UK) and/or Europe (EU). |
| Clinical Investigation Type | Retrospective-prospective, multi-center, non-randomized, unblinded, post-market study to evaluate the long-term performance and safety of AtriClip® FLEX-V LAA and PRO•V LAA Exclusion devices for exclusion of the left atrial appendage of the heart during concomitant cardiac procedures. |
| AtriCure Medical Advisor | Sydney Gaynor Medical Director of Clinical Education, Clinical AtriCure, Inc. 7555 Innovation Way, Mason, OH 45040 M. 513-560-5974 SGaynor@atricure.com |
| Sponsor | Pam Simons VP, Clinical Affairs AtriCure, Inc. 7555 Innovation Way, Mason, OH 45040 O. 763-260-5267 PSimons@atricure.com |
| Electronic Data Capture<br>Software | Clindex® |
| Core Laboratories | NYU Langone Health, NY |
| Independent Physician Adjudicator(s) | To be Determined |
| Protocol Author | Rebecca Ikura, Senior Clinical Project Manager |

Protocol Number: CP-2021-03 Protocol Name: V-CLIP Study Version: Rev B; Oct 15, 2021 



#### **CONFIDENTIALITY STATEMENT**

The information in this document contains trade secrets and commercial information that are privileged or confidential to AtriCure, Inc. and may not be disclosed unless such disclosure is required by federal or state law or regulations. Subject to the foregoing, this information may be disclosed only to those persons involved in the trial who have a need to know, but all such persons must be instructed not to further disseminate this information to others. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

# **SPONSOR SIGNATURE PAGE**

| Trial Name | VCLIP Study | | |
|---|---|---|---|
| Trial Number: | CP-2021-03 | | |
| Title: | Long-Term Follo | w-Up on LAA Exclusion usir | ng AtriClip |
| Test Articles: | AtriCure AtriClip@ | 3 LAA Exclusion system cor | mprised of: |
| | • Flex-V (ACHV) | and PRO•V | |
| Approvals: | | | |
| Electronic approvals obtained this document. | via AtriCure's Qualit | y System (Master Control) are | located at the end of |
| See MasterControl | | See MasterControl | |
| Pam Simons VP Clinical Affairs AtriCure, Inc. See MasterControl | Date | Sydney Gaynor, MD Medical Director of Clinical E AtriCure, Inc. See MasterControl | Date<br>ducation, Clinical |
| | Date | Yashasvi Awasthi | Date |
| Dennis Hong, JD, RAC<br>VP, Regulatory Affairs | Date | VP Global Scientific Affairs a | |
| AtriCure, Inc. | | AtriCure, Inc. | and Evidence endlegy |
| See MasterControl | | See MasterControl | <b>5</b> / |
| Nfii Ndikintum | Date | Jesse Sheridan | Date |
| VP Clinical Affairs & Biometrics | S | Pr. Clinical Database Program | mmer |


AtriCure, Inc.

AtriCure, Inc.

See MasterControl
Rebecca Ikura

Sr. Clinical Project Manager


Form-582.B

Date

AtriCure, Inc.



## SITE INVESTIGATOR PROTOCOL SIGNATURE PAGE / INVESTIGATOR AGREEMENT

I have read, understood, and agree to:

- Ensure that the requirements for obtaining informed consent are met
- Conduct the trial in accordance with this protocol, including applicable local/state laws and regulations
- Provide a copy of the Financial Disclosure form that summarizes financial interest in AtriCure. Inc.
- Complete all Case Report Forms and study documentation, and relevant assessments (as required) promptly to the Sponsor, AtriCure, Inc., or its authorized representatives
- Adhere to the publication policy of AtriCure, as stated in the Clinical Study Agreement, for data collected during this trial
- Ensure that all associates, colleagues, and employees of AtriCure assisting in the conduct of the trial(s) are informed of their obligations in meeting the above commitments
- Propose to the sponsor any appropriate modification(s) of the protocol or investigational device, or of the use of the investigational device

I will ensure that the IRB/EC review complies with governmental requirements and will be responsible for the initial and continuing review and approval of the clinical investigation. I also agree to promptly report to the IRB/EC all changes in the research activity and all unanticipated problems involving risks to human subjects or others. Additionally, I will not make any changes in the research without sponsor and IRB/EC approval of an amended protocol, except where necessary to eliminate apparent immediate hazards to human subjects.

I have read and agree to adhere to the clinical investigation plan and all regulatory requirements applicable in conducting this clinical investigation.

Site Principal-Investigator / Sub-Investigator

| Printed name: |
|---------------|
| Signature: |
| Date: |

Please return the signed form to your site assigned CRA

AtriCure, Inc. (Sponsor) 7555 Innovation Way Mason, Ohio 45040

Protocol Number: CP-2021-03 
Protocol Name: V-CLIP Study

Version: Rev B; Oct 15, 2021 Form-582.B



# **VCLIP PROTOCOL SYNOPSIS**

| Regulatory<br>Classification | Post-Market Study |
|---|---|
| Indication | The AtriCure AtriClip LAA Exclusion system is indicated for the exclusion of the heart's left atrial appendage, performed under direct visualization and in conjunction with other cardiac surgical procedures. |
| Clinical<br>Investigation<br>Name and<br>Number | VCLIP Post-Market Study<br>CP-2021-03 |
| Title | Long-Term Follow-Up on LAA Exclusion using AtriClip |
| Objective(s) | The objective of this trial is to evaluate the long-term performance and safety of the AtriClip FLEX-V and PRO•V LAA Exclusion devices for exclusion of the left atrial appendage. |
| Device(s) Under | AtriCure AtriClip LAA Exclusion system comprised of: |
| Investigation | • Flex-V (ACHV) and PRO•V |
| Rationale | The study proposed herein is to gather clinical data on the long-term performance and safety of the AtriClip FLEX-V and PRO•V LAA Exclusion devices. Data from this study may be used for submission to regulatory authorities in the US, Europe, China and other geographies as needed, as well as for publication purposes. |
| Number of Subjects/Sites | Up to 170 subjects will be enrolled at up to 20 sites in the US, UK and/or EU. |
| Clinical<br>Investigation<br>Design | Retrospective-prospective, multi-center, non-randomized, unblinded, post-market study to evaluate the long-term performance and safety of AtriClip FLEX-V LAA and PRO•V LAA Exclusion devices for exclusion of the left atrial appendage of the heart during cardiac procedures. |
| Subject<br>Population | Subjects who have undergone designated non-emergent, cardiac surgical procedure(s), received an AtriClip implant (with devices under investigation) and who are willing to return for follow-up chest imaging to ascertain Left Atrial Appendage (LAA) exclusion will be eligible to participate based upon the inclusion and exclusion criteria. |
| | Subjects who had received chest imaging for other reasons, and if the imaging includes pertinent information to verify LAA exclusion, will also be eligible to participate if they meet eligibility criteria. |




| Justification of Sample Size and | A minimum sample size of 170 subjects is required to evaluate the primary performance of LAA exclusion at 12-months using the following assumptions: |
|---|---|
| Performance Goal | Test basis: exact test for one proportion |
| | 1-sided alpha: 0.025 |
| | Power: 92% |
| | Performance Goal: 80% |
| | Expected closure rate: 90% |
| | Expected attrition rate: 16% |
| | Based on these assumptions, a minimum of 143 subjects are required before accounting for attrition. To account for an estimated attrition of 16% for subjects that consent but miss the imaging during follow-up, a total of 170 subjects will need to be enrolled. |
| | Performance goal: The 12-month LAA closure rate (No leak) for contemporary devices ranges from 66 % - 89.5%. In-line with these rates, a PG of 80% is proposed for this study. |
| | In addition, based on a performance goal of 10.5% for safety at 30-days post AtriClip implantation, expected SAE rate of up to 5%, the sample size provides 85.4% power to demonstrate primary safety success. |
| Inclusion Criteria | <ol> <li>Subject is greater than or equal to 18 years of age.</li> <li>Subject who received the AtriClip FLEX-V or PRO•V implant during a non-emergent cardiac surgical procedure</li> <li>Subject is willing and able to provide written informed consent</li> <li>Subject is willing and able to return for scheduled follow-up visit and imaging (CTA or TEE)</li> </ol> |
| Exclusion Criteria | <ol> <li>Inability, unwillingness, or contraindication to undergo TEE or CTA imaging</li> <li>Subjects who are pregnant or breast feeding</li> <li>Subjects with active COVID-19 infection</li> </ol> |
| Subject Follow-up | Treated subjects will be assessed for long-term performance and safety at 12-months or greater post-procedure (i.e., the last follow-up visit). |
| Primary<br>Endpoint(s) | Primary Performance Endpoint 1. Left Atrial Appendage exclusion defined as absence of residual communication (no leaks) between the left atrium (LA) and the LAA as assessed by CTA or TEE imaging at the last follow-up visit. The images will be reviewed by an independent core lab using a standardized imaging protocol. |
| | Primary Safety Endpoint |




| | <ol> <li>Incidence of the following serious adverse events within 30-days, if related to the device and/or implant procedure: <ul> <li>Death</li> <li>Major Bleeding (BARC 3 and above)</li> <li>Surgical site infection</li> <li>Pericardial effusion requiring intervention</li> <li>Clinical diagnosis of myocardial infarction</li> </ul> </li> <li>The safety events will be adjudicated by an independent medical monitor (cardiac surgeon).</li> </ol> |
|---|---|
| Secondary<br>Endpoints | <ol> <li>A residual LAA neck ≤10 mm as assessed by CTA or TEE imaging at the last follow-up visit</li> <li>Device or procedure related SAEs through the last follow-up visit</li> <li>These data will be descriptively summarized by reporting the counts and percentages of each event reported.</li> </ol> |




# **TABLE OF CONTENTS**

| VCL | IP POST-MARKET STUDY | 1 |
|---|---|---|
| | DNSOR SIGNATURE PAGE | |
| VCL | IP PROTOCOL SYNOPSIS | 4 |
| 1 | INTRODUCTION | 12 |
| 1. | | |
| | 1.1.1 Background | 12 |
| | 1.1.2 Rationale for Conducting this Clinical Investigation | 12 |
| 2 | CLINICAL INVESTIGATION OVERVIEW | |
| 2. | 1 Clinical Investigation Objective | 13 |
| 2.: | 2 Investigational Device(s) To Be Used in the Clinical Investigation | 13 |
| 2.: | 2.1 Name of the Device(s) Under Investigation | 13 |
| 2. | 2.2 Indication for Use | |
| 2. | 2.3 Description of the Device(s) Under Investigation | |
| 2. | 2.4 Device Handling | 13 |
| 3 | CLINICAL INVESTIGATION DESIGN | 13 |
| 3. | 1 Clinical Investigation Procedures and Follow-up Schedule | 14 |
| 3. | 2 Measures Taken to Avoid and Minimize Bias | 14 |
| 3. | | |
| 4 | ENDPOINTS | 15 |
| 4. | 1 Primary Safety Endpoint | 15 |
| 4. | 2 Primary Performance Endpoint | 15 |
| 4. | 3 Secondary Endpoint | 16 |
| 4. | 4 Descriptive Endpoint(s) or Additional Data | 16 |
| 5 | SUBJECT SELECTION AND WITHDRAWAL | 16 |
| 5. | 1 Subject Population | 16 |
| 5. | 2 Subject Screening and Informed Consent | 16 |
| 5. | 2.1 Subject Screening | 16 |
| 5. | 2.2 Informed Consent | |
| 5. | 2.2.1 Special Circumstances for Informed Consent | 18 |
| 5. | 3 Eligibility Criteria | 18 |




| | 5.3.1 | General Eligibility Criteria | 18 |
|---|---|---|---|
| | 5.3.2 | Inclusion Criteria | 18 |
| | 5.3.2. | 1 General Inclusion Criteria | 18 |
| | 5.3.3 | Exclusion Criteria | 19 |
| | 5.3.3. | 1 General Exclusion Criteria | 19 |
| | 5.4 | Subject Enrollment | 19 |
| | 5.4.1 | Historically Under-Represented Demographic Subgroups | 19 |
| | 5.5 | Subject Withdrawal | |
| | 5.6 | Number of Subjects | 21 |
| | 5.7 | Total Expected Duration of the Clinical Investigation | |
| 6 | TRE | EATMENT AND EVALUATION OF ENDPOINTS | 21 |
| | 6.1 | Study Eligibility | |
| | 6.2 | Retrospective Follow-up Assessments | 21 |
| | 6.2.1 | Baseline (within 30 days prior to index procedure) | 21 |
| | 6.2.3 | 30-days Post-Procedure Visit, if done (+/- 7 days) | 22 |
| | 6.3 | Prospective Follow-up Assessments | 22 |
| | 6.3.1 | 12-Month Post-Procedure Visit (≥ 12months) | |
| | 6.3.2 | Study Exit | |
| | 6.3.3 | Schedule of Events | 23 |
| | 6.4 | Requirement for Clinical Laboratories | 24 |
| 7 | AD\ | VERSE EVENTS | 24 |
| | 7.1 | Definition | 24 |
| | 7.1.1 | Adverse Event | 24 |
| | 7.1.2 | Serious Adverse Event | 24 |
| | 7.1.3 | Device Deficiency/Device Malfunction | 25 |
| | 7.2 | Pre-Existing Conditions Versus Adverse Events | 25 |
| | 7.3 | Severity of Adverse Events | 25 |
| | 7.4 | Device Relationship | 26 |
| | 7.4.1 | Unanticipated (Serious Adverse) Device Effect [U(S)ADE] | 27 |
| | 7.5 | Adverse Event and Device Deficiency/Device Malfunction Reporting | 27 |
| | 7.5.1 | AE/ADE/UADE Reporting | 27 |
| | 7.5.2 | SAE/USADE Reporting | 27 |
| | 7.5.3 | Device Deficiency/Malfunction Reporting | 28 |




| | 7.5.4 | Adverse Event Reporting to Country Regulatory Authorities by the Sponsor | 29 |
|---|---|---|---|
| | 7.6 | Expected Morbidity/Procedural Complications Reporting | 29 |
| | 7.7 | Product Complaints | 30 |
| | 7.7.1 | Reporting Product Complaints | 30 |
| | 7.7.2 | Reporting Product Complaints with Non-Investigational Device Products | 31 |
| | 7.7.3 | Non-AtriCure Product Complaints | 31 |
| | 7.7.4 | Reporting Product Complaints for Global Compliance | 31 |
| 8 | STA | ATISTICAL CONSIDERATIONS | 31 |
| | 8.1 | Analysis Populations | 31 |
| | 8.2 | Statistical Analyses | 31 |
| | 8.2.1 | Primary Performance Endpoint Analysis | 32 |
| | 8.2.2 | Primary Safety Endpoint Analysis | 32 |
| | 8.2.3 | Secondary Endpoint Analyses | 32 |
| | 8.2.4 | Long-Term Safety Analyses | 33 |
| | 8.3 | Sample Size Calculation and Assumptions | 33 |
| | 8.4 | Timing of Analysis | 34 |
| | 8.5 | Subgroup Analysis | |
| | 8.6 | Multiplicity | |
| | 8.7 | Pooling Strategy | 34 |
| | 8.8 | Procedures for Accounting for Missing Data | 34 |
| | 8.9 | Statistical Criteria for Termination | 34 |
| | 8.10 | Success Criteria | 34 |
| | 8.11 | Deviations from Statistical Plan | 34 |
| 9 | DIR | ECT ACCESS TO SOURCE DATA/DOCUMENTS | 34 |
| 1 | 0 C | UALITY CONTROL AND QUALITY ASSURANCE | 35 |
| | 10.1 | Selection of Clinical Sites and Investigators | 35 |
| | 10.2 | Clinical Investigation Finances and Agreements | 35 |
| | 10.3 | Protocol Amendments | 35 |
| | 10.4 | Training | 35 |
| | 10.4.1 | Site Training | 35 |
| | 10.5 | Monitoring | 36 |
| | 10.6 | Protocol Deviations | 36 |
| | 10.7 | Quality Assurance Audit | 37 |




| 10.8 | B Committees | .37 |
|---|---|---|
| 10.8 | 3.1 Study Oversight Committee | .37 |
| 10.8 | 3.2 Publications Committee | .38 |
| 10.8 | 3.3 Independent Physician Adjudicator (IPA) | .38 |
| 11 | DATA HANDLING AND RECORD KEEPING | .38 |
| 11.1 | Protection of Personally Identifiable Information | .39 |
| 11.2 | 2 Data Management Plan | 40 |
| 11.3 | Source Documentation | 40 |
| 11.4 | Case Report Form Completion | 40 |
| 11.5 | Record Retention | 40 |
| 11.6 | 5 | |
| 12 | ETHICAL CONSIDERATION | .41 |
| 12.1 | Institutional Review Board/Medical Ethics Committee Review and Approval | 41 |
| 13 | CLINICAL INVESTIGATION CONCLUSION | 42 |
| 14 | PUBLICATION POLICY | |
| 15 | RISK ANALYSIS | |
| 15.1 | Anticipated Clinical Benefits | 42 |
| 15.2 | Profeseeable Adverse Events and Anticipated Adverse Device Effects | 42 |
| 15.3<br>Risk | Residual Risks Associated with the Device Under Investigation, as Identified in the<br>VQuality Management Report | .43 |
| 15.4 | | |
| 15.5 | Steps Taken to Control or Mitigate Risks | .43 |
| 15.6 | Risk to Benefit Rationale | .43 |
| APPE | NDIX I: REFERENCES | .44 |
| APPE | NDIX II: ABBREVIATIONS AND ACRONYMNS | .45 |
| APPE | NDIX III: DEFINITIONS | .47 |
| APPE | NDIX IV: FORSEEABLE ADVERSE EVENTS | .58 |
| APPE | NDIX V: INFORMED CONSENT FORM | .60 |
| APPE | NDIX VI: SITE CONTACT INFORMATION | .61 |
| APPE | NDIX VII: REVISION HISTORY | .62 |



#### **COMPLIANCE STATEMENT**

This clinical investigation will be conducted in accordance with this Clinical Investigation Plan, the Declaration of Helsinki, applicable Good Clinical Practices and regulations (e.g., US 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 812 and OUS ISO14155:2020) and any other appropriate local regulations(s). The most stringent requirements, guidelines or regulations must always be followed. The conduct of the clinical investigation will be approved by the appropriate Institutional Review Board (IRB)/Ethics Committee (EC) of the respective investigational site and by the applicable regulatory authorities prior to study enrollment.

This clinical investigation will be financed by AtriCure. Investigational sites will be compensated by AtriCure for participation in the clinical investigation per the conditions of Clinical Trial Agreement (CTA) between the Sponsor and the Investigational site.




#### 1 INTRODUCTION

This clinical investigation will be conducted in accordance with this Clinical Investigational Plan (CIP), also referred to herein as the "Protocol". All investigators involved in the conduct of the clinical investigation will be qualified by education, training, or experience to perform their tasks and the training will be documented appropriately. The investigator will create and maintain source documents throughout the clinical investigation and make them available as requested during monitoring visits or audits, as well as maintain documentation of the type and location of these source documents. The investigator will also determine the cause and implement appropriate corrective and preventative actions to address any significant noncompliance that arise during the conduct of the study/trial.

# 1.1 Background and Rationale

# 1.1.1 Background

Exclusion or excision of the left atrial appendage (LAA) has been performed since the late 1940s. Left atrial appendage suture-enabled exclusion/excision is intended to prevent thrombi that are developed in the heavily trabeculated LAA from migrating outside of the LAA. In patients with AF >90% of thrombi are generated in LAA. These thrombi can dislodge from left atrium and migrate to other parts of the body and can cause ischemic events hence it is important to close or exclude LAA to avoid thrombus from escaping.

Various surgical techniques include: epicardial suture occlusion (ligation), endocardial suture occlusion, stapling, and surgical excision. These techniques are associated with incomplete LAA closure rates of 40% to 60% and the technique can be difficult, adding significant cross clamp time.<sup>1-6</sup>

Results of the randomized control pilot Left Atrial Appendage Occlusion Study (LAAOS) were reported by Healy et al.<sup>7</sup> The LAAOS study assessed the safety and efficacy of LAA exclusion performed at the time of coronary artery bypass grafting (CABG) using sutures or a stapling device. It was shown that among patients having a postoperative transesophageal echocardiogram (TEE), complete exclusion of the LAA was achieved in 45% of cases using sutures and in 72% using a stapler. Given the low rate of exclusion with these techniques there is a need to exclude LAA using the device that provides an improved rate of closure.

#### 1.1.2 Rationale for Conducting this Clinical Investigation

This study is proposed herein is to gather clinical data on the long-term performance and safety of the AtriClip FLEX-V and PRO•V LAA Exclusion devices.

Data from this study may be used for submission to regulatory authorities in the US, Europe, China and other geographies as needed, as well as for publication purposes.




#### 2 CLINICAL INVESTIGATION OVERVIEW

# 2.1 Clinical Investigation Objective

The primary objective of this study is to demonstrate the long-term performance and safety of the AtriClip FLEX-V and AtriClip PRO•V devices to successfully exclude the LAA with absence of residual communication between the LA and the LAA at the last follow-up visit post AtriClip implant.

# 2.2 Investigational Device(s) To Be Used in the Clinical Investigation

The subject device for this study will be the AtriCure AtriClip LAA Exclusion system, which has been cleared under the 510 (k) process by the FDA and is approved in the UK and EU for commercial use. It is therefore not an investigational device.

The AtriCure AtriClip LAA Exclusion system is comprised of:

• Flex-V (ACHV) and PRO•V

## 2.2.1 Name of the Device(s) Under Investigation

Please refer to the IFU for additional information regarding the device used in this clinical investigation.

#### 2.2.2 Indication for Use

The AtriCure AtriClip LAA Exclusion system is indicated for the exclusion of the heart's left atrial appendage (LAA), performed under direct visualization and in conjunction with other cardiac surgical procedures.

Direct visualization in this context, requires that the surgeon was able to see the heart directly, with or without assistance from a camera, endoscope, etc., or any other appropriate viewing technology.

#### 2.2.3 Description of the Device(s) Under Investigation

Please refer to the IFU for additional information regarding the device used in this clinical investigation.

## 2.2.4 Device Handling

Subjects enrolled in this study will already have been treated with commercial devices; therefore, device accountability is not required.

#### 3 CLINICAL INVESTIGATION DESIGN

This is a retrospective-prospective, multi-center, non-randomized, unblinded, post-market study sponsored by AtriCure, Inc. This study will evaluate the long-term performance and safety of the AtriClip FLEX-V LAA and PRO•V LAA Exclusion Systems for exclusion of the LAA of the heart during concomitant cardiac procedures. Specifically, the implanted clip (AOD2) for both the AtriCure FLEX-V and PRO•V devices will be evaluated. This study will be conducted in the US, EU and UK under a single protocol approved by an IRB/EC for each site prior to study enrollment at the site. The Principal Investigators (PIs) acknowledges the responsibilities described in the Protocol Signature Page.




The PIs at the sites are cardiac surgeons, qualified by education, experience, and training to assume responsibility for the conduct of this study. Up to 20 sites will participate in the study.

Up to 170 subjects will be enrolled as part of the study. Treated subjects will be assessed for long-term performance and safety at 12-months or greater post-procedure.

An independent Core Lab will be utilized for evaluation of the CTA and TEEs. All prospective assessments should be performed in accordance with the Core Labs recommended protocol.

An Electronic Data Capture (EDC) system will be utilized by study site personnel to transfer study data from source records (medical records and/or source document worksheets) onto common electronic case report forms (eCRFs). This system is a web-based, secure electronic software application, (Clindex®), developed and maintained by Fortress Medical Systems in a manner that is compliant with national and international GCP data protection/data privacy and electronic record/electronic signature (e.g., 21 CFR Part 11) regulatory requirements.

Adverse Events and medical device performance issues (for medical devices used during the procedure), including potential and actual device-related adverse events, certain malfunctions and user errors suspected to be associated with the use of a Food and Drug Administration (FDA) regulated drug, biologic, medical device or dietary supplement used during the course of this study will be reported by the PI to applicable authorities including the: 1) Sponsor (AtriCure); 2) IRB/EC; 3) respective manufacturer(s); and/or 4) FDA via MedWatch Online Voluntary Reporting Process or Medical Device Reporting as appropriate.

Critical decisions related to the design and execution of the study will be managed by the National PI and AtriCure's Medical Advisor.

The clinical investigation has been designed to involve as little pain, discomfort, fear, and any other foreseeable risk as possible for subjects. Refer to the Risks Analysis section of this protocol for details.

#### 3.1 Clinical Investigation Procedures and Follow-up Schedule

Clinical investigation sites that have treated subjects with either the AtriClip FLEX-V or PRO•V device will be approached to determine if they are resourced and willing to consent subjects treated at least 12-months post procedure for LAA closure imaging (CTA or TEE). The follow-up assessment data will be entered into the electronic data system developed for the study.

Documentation and reason for screen failure (i.e., inability to consent, refused consent, did not meet inclusion exclusion criteria, death or major morbidity such as stroke, etc. will be secured on a screening log within EDC.

## 3.2 Measures Taken to Avoid and Minimize Bias

This is a single-arm study. All enrolled subjects would have been treated with either the AtriClip FLEX-V or PRO•V device. Study data will be monitored against relevant source documents. An




independent physician will adjudicate the SAEs reported in the study and LAA closure imaging will also be adjudicated by a core lab. Furthermore, to mitigate temporal bias, enrollment in the trial will be based on random selection of treated subjects. The sequence with which treated subjects will be screened and invited to participate in the trial will be randomly generated by the sponsor and provided to each site.

#### 3.3 Suspension or Early Termination of the Clinical Investigation

The Sponsor reserves the right to discontinue the clinical investigation at any stage with suitable written notice to the investigator. Possible reason(s) may include, but are not limited to:

A Study Oversight Committee (e.g., National PI(s) & AtriCure Medical Advisor)
makes a recommendation to stop or terminate the clinical investigation.

Should the clinical investigation be discontinued by the Sponsor, subjects will be followed per routine hospital standard of care with device-related AEs reported to the Sponsor as per vigilance/commercial reporting requirements. All applicable clinical investigation documents shall be subject to the same retention policy as detailed in [Section 11.5] of the Protocol.

A Principal Investigator, IRB/EC or regulatory authority may suspend or prematurely terminate participation in the clinical investigation at the investigational site(s) for which they are responsible. The investigators will follow the requirements specified in the Clinical Trial Agreement.

If the Sponsor suspends or prematurely terminates the clinical investigation at an individual site in the interest of safety, the Sponsor will inform all other sites and Principal Investigators.

If suspension or premature termination occurs, the Principal Investigator or authorized designee will promptly inform the enrolled subjects at his/her site, if appropriate, and return subjects to their standard of care medical treatment.

# 4 **ENDPOINTS**

# 4.1 Primary Safety Endpoint

This endpoint is defined as the incidence of the following serious adverse events (SAEs) within 30-days, if related to the device and/or implant procedure:

- Death
- Major Bleeding (BARC 3 and above)
- Surgical site infection
- Pericardial effusion requiring intervention
- Clinical diagnosis of myocardial infarction

Refer to Appendix III for definitions of each of the events.

#### 4.2 Primary Performance Endpoint

This endpoint includes LAA exclusion defined as absence of residual communication (i.e. no leak) between the left atrium and the LAA, assessed by CTA or TEE imaging at the last follow-up visit.




#### 4.3 Secondary Endpoint

Key Secondary Endpoints include:

- 1. A residual LAA neck ≤10 mm as assessed by CTA or TEE imaging at the last follow-up visit
- 2. Device or procedure related SAEs through the last follow-up visit

These data will be descriptively summarized by reporting the counts and percentages of each event reported.

# 4.4 Descriptive Endpoint(s) or Additional Data

If necessary, additional analyses and endpoints will be defined in a separate Statistical Analysis Plan (SAP) prior to database lock.

## 5 SUBJECT SELECTION AND WITHDRAWAL

## 5.1 Subject Population

This clinical investigation will enroll subjects who have undergone designated non-emergent, cardiac surgical procedure(s) and received an AtriClip implant (with the devices under investigation), and who are willing to return for follow-up chest imaging to ascertain LAA exclusion. Subjects must meet all eligibility criteria and provide written informed consent prior to collection of study data.

Subjects who had received chest imaging for other reasons and the image includes pertinent information to verify LAA exclusion, will also be eligible to participate if they meet eligibility criteria.

# 5.2 Subject Screening and Informed Consent

#### 5.2.1 Subject Screening

Potential patients presenting at the clinical sites will be fully informed about the clinical investigation, following the established Informed Consent process (described in [Section 5.2.2]).

Subjects must be screened for clinical investigation eligibility by a member of the site's clinical investigation team trained to the protocol, and if applicable will be entered into a site-specific screening log.

In case the subject does not meet all inclusion criteria or meets any of the exclusion criteria, the subject is considered a screening failure. The Principal Investigator or the delegated clinical investigation personnel will record the reasons for screen failure (e.g., inability to consent, refusal to consent, did not meeting inclusion/exclusion criteria, death or major morbidity (e.g., stroke) etc. on a screening log within the EDC as required.




Patients meeting general inclusion criteria and no exclusion criteria will be asked to sign an Informed Consent form if they wish to participate in the clinical investigation. These patients will also be entered into the screening log.

Subject data will be collected following enrollment into the clinical investigation and will be based on random selection of treated subjects.

#### **5.2.2 Informed Consent**

The Informed Consent Form (ICF) must have the approval of the IRB or favorable opinion of the EC. While some institutions may request modification of the ICF to satisfy specific institutional requirements, the use of a modified or unique ICF is permitted if it meets the requirement of 21 CFR Part 50 and ISO 14155:2020 and is approved by the Sponsor.

The Investigator or his/her authorized designee will conduct the Informed Consent process, as required by applicable regulations and the center's IRB/EC. This process will include a verbal discussion with the subject on all aspects of the clinical investigation that are relevant to the subject's decision to participate, such as details of clinical investigation procedures, anticipated benefits, and potential risks of clinical investigation participation. Subjects must be informed about their right to withdraw from the clinical investigation at any time and for any reason without sanction, penalty or loss of benefits to which the subject is otherwise entitled. Withdrawal from the clinical investigation will not jeopardize their future medical care or relationship with the investigator.

During the discussion, the Principal Investigator or his/her authorized designee will avoid any improper influence on the subject and will respect subject's legal rights. Financial incentives will not be given to the subject. Subjects may be compensated for time and travel directly related to the participation in the clinical investigation. The subject shall be provided with the Informed Consent form written in a language that is understandable to the subject and has been approved by the center's IRB/EC. The subject shall have adequate time to review, ask questions, and consider participation. The Principal Investigator or his/her authorized designee will make efforts to ensure that the subject understands the information provided. If the subject agrees to participate, the Informed Consent form must be signed and dated by the subject and thereafter by the person obtaining the consent prior to any clinical investigation-specific procedures. The signed original will be filed in the subject's hospital or research charts, and a copy will be provided to the subject.

Failure to obtain Informed Consent from a subject prior to clinical investigation enrollment should be reported to Sponsor within 5 working days and to the reviewing center's IRB/EC according to the IRB's/ EC's reporting requirements.

If, during the clinical investigation, new information becomes available that can significantly affect a subject's future health and medical care, the Principal Investigator or his/her authorized designee (if applicable) will provide this information to the subject. If relevant, the subject will be asked to confirm their continuing Informed Consent in writing.




The ICF will clearly stipulate that the duration of the study is approximately 1.5 years, and the implications of this commitment will be reviewed and discussed with the subjects prior to enrollment in the study.

#### 5.2.2.1 Special Circumstances for Informed Consent

For eligible subjects in the U.S. an authorization for use and disclosure of the subject's protected health information, in accordance with the Health Insurance Portability and Accountability Act (HIPAA), must be obtained from the subject or their legally acceptable representative.

For subjects outside of the U.S. (OUS), a separate GDPR consent may be required if not already included within the ICF.

In addition,

- Individuals under the age of 18 or age of legal consent are excluded from the study population.
- Pregnant or breastfeeding women are excluded from the study population.

Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population.

For individuals unable to read or write, Informed Consent will be obtained through a supervised oral process. An independent witness will be present throughout the Informed Consent process. The written Informed Consent form and any other information will be read aloud and explained to the prospective subject or his/her legally acceptable representative and either will sign and personally date the Informed Consent form. The witness will also sign and personally date the Informed Consent form attesting that the information was accurately explained, and that Informed Consent was freely given.

#### 5.3 Eligibility Criteria

#### 5.3.1 General Eligibility Criteria

Assessment for general eligibility criteria is based on medical records at the site and interview with a candidate subject. Subjects must meet ALL of the inclusion criteria to be considered for the clinical investigation. If ANY of the exclusion criteria are met, the subject is excluded from the clinical investigation and cannot be enrolled.

# 5.3.2 Inclusion Criteria

#### 5.3.2.1 General Inclusion Criteria

All subjects recruited for study participation must meet all of the following inclusion criteria to be enrolled in the study:

- 1. Subject is greater than or equal to 18 years of age
- 2. Subject who received the AtriClip FLEX-V or PRO•V implant during a non-emergent cardiac surgical procedure
- 3. Subject is willing and able to provide written Informed Consent




4. Subject is willing and able to return for scheduled follow-up visit and imaging (CTA or TEE)

#### 5.3.3 Exclusion Criteria

#### 5.3.3.1 General Exclusion Criteria

Potential subjects required for study participation must not meet any of the following exclusion criteria to be enrolled in the study:

- 1. Inability, unwillingness, or contraindication to undergo TEE or CTA imaging
- 2. Subjects who are pregnant or breast feeding
- 3. Subjects with active COVID-19 infection.

## 5.4 Subject Enrollment

Subjects will be provided the IRB/EC approved ICFs and will have the opportunity to read, understand, and have their questions answered prior to signing the ICFs. If the subject agrees to participate in the study and signs consent, the ICF process will be completed. The subject must sign and date the ICF prior to collection of study data. The person reviewing the ICF with the subject will also sign and date the ICFs. The subject will be given a copy of the signed ICF for their personal records.

Upon entering subject enrollment information into Clindex, each subject will be assigned a unique identification (ID) number sequentially in ascending order. All subjects who sign the ICFs will be documented in a Screening and Enrollment Log. For subjects who sign the ICF but are ineligible to participate, minimum baseline characteristics (e.g., age, gender, race, screening date and screen failure reason, etc.) will be captured in Clindex.

A subject is considered enrolled in the clinical investigation from the moment the subject provides written Informed Consent and has been confirmed to meet all inclusion criteria and none of the exclusion criteria.

# 5.4.1 Historically Under-Represented Demographic Subgroups

AtriCure will take the following steps to ensure adequate representation of women and racial or ethnic minorities in this clinical investigation:

- as appropriate and necessary, AtriCure will train sites on the importance of recruiting and retaining subjects in the clinical investigation
- approach sites without bias or consideration for specific demographic subgroups
- have Informed Consent materials in alternative languages and will work with sites and IRBs/ECs on recruitment materials.

# 5.5 Subject Withdrawal

Each enrolled subject shall remain in the clinical investigation until completion of the required follow-up period; however, a subject's participation in any clinical investigation is voluntary and the subject has the right to withdraw at any time without penalty or loss of benefit. Conceivable reasons for discontinuation may include, but not be limited to, the following:

- Subject death
- Subject voluntary withdrawal




- Subject lost-to follow-up as described below
- Subject's follow-up is terminated due to site/study termination

The Sponsor must be notified by the site of the reason(s) for subject discontinuation and record a reason for termination in the case report form (CRF). Investigators must also report this to their respective IRB/EC as defined by their institution's procedure(s).

#### Investigator Decision

If the subject experiences an adverse event and the Principal Investigator or Medical Advisor believes it is in their best interest to discontinue participation in the study, they will be withdrawn from the study.

## Lost to follow-up

If the subject misses their scheduled follow-up and the attempts at contacting the subject detailed below are unsuccessful, then the subject is considered lost-to-follow-up. Site personnel shall make all reasonable efforts to locate and communicate with the subject (and document these efforts in the source documents), including the following, at each contact time point:

- A minimum of two telephone calls on different days and times should be recorded in the source documentation, including date, time and initials of site personnel trying to make contact.
- If these attempts are unsuccessful, a letter (certified if applicable) should be sent to the subject.

#### Withdrawal of consent

The subject withdraws consent for participation in the study. Any method of contact with the subject in which they state they no longer want to participate in the study specific activities constitutes withdrawal of consent. When possible, the reason for withdrawal will be documented.

<u>Death:</u> Subject expires after enrollment into the study.

## Site Termination or Study Termination

A site or the study may be terminated. When this occurs all subjects at the site will be withdrawn and documented as early termination. Reasons for site or study termination may include, but are not limited to the following:

- Administrative concerns (e.g., inadequate subject enrollment, Investigator/institution non-compliance, change of business strategy, etc.);
- Safety issues, including those due to non-compliance, which substantially affect the risk to benefit ratio of the study subjects at a site or for the study as a whole;
- Regulatory body mandate(s).

# Other (which may include)

- Protocol deviation, noncompliance, or violation;
- Investigator/Sponsor recommendation;

#### Follow-up for Early Terminated Subjects




Given the nature of the study procedures, there are situations where subjects may terminate from the study early that are not described above. No additional follow—up will be required or data recorded from subjects once withdrawn from the clinical investigation, except for the status (deceased/alive). The investigator can use existing data and ask for the subject's permission to collect follow-up data about his/her status/condition including information about device clinical performance or safety. If permission is obtained, the relevant data shall be included in the clinical investigation report.

# 5.6 Number of Subjects

Up to 170 subjects will be enrolled at up to 20 sites in the US, UK and/or EU.

# 5.7 Total Expected Duration of the Clinical Investigation

The expected duration of the study is approximately 21 months. Enrollment will be closely monitored and AtriCure will work directly with the sites to clearly understand the enrollment challenges they might be facing, retrain as needed and pursue other strategies to address any enrollment lapse. Subjects will be exited from the trial at the conclusion of their primary performance follow-up visit occurring at least 12-months post-procedure.

## 6 TREATMENT AND EVALUATION OF ENDPOINTS

## 6.1 Study Eligibility

All subjects recruited for study enrollment must meet all study enrollment criteria prior to being enrolled in the study. The clinical investigation site will review all subjects treated with either the AtriClip FLEX-V or PRO•V device. Once the initial chart review indicates that the subject meets the study inclusion / exclusion criteria, the subject will be approached for their interest in the study, including willingness to return for their follow-up visit.

#### 6.2 Retrospective Follow-up Assessments

Once the subject is consented, the following data will be collected by reviewing the subjects' medical records retrospectively. For retrospective visits that fall outside of the required windows, please refer to section 10.6 (Protocol Deviations).

## 6.2.1 Baseline (within 30 days prior to index procedure)

- Inclusion/Exclusion criteria
- Demographic information (Age, Sex, Race, Ethnicity)
- Review of Medical and Cardiac history, including CHADS, CHADSVASC, and HASBLED scores, if available
- Vital Signs (BMI, Blood Pressure, Heart Rate)
- NYHA Classification
- Medication history (e.g., Anticoagulants, antihypertensives, etc.,). Medication information should include:
  - o Name
  - Dosage with units

# 6.2.2 Start Index Procedure




- Evaluation of any adverse events AEs/SAEs that occur up to discharge
- Concomitant surgical procedure
- Intra-op TEE pre-clip placement for thrombus, if done (e.g., LA Size)

# 6.2.3 30-days Post-Procedure Visit, if done (+/- 7 days)

- NYHA Classification
- Evaluation of any AEs/SAEs

# 6.3 Prospective Follow-up Assessments

#### 6.3.1 12-Month Post-Procedure Visit (≥ 12months)

Subjects will be asked to return to the clinic for a final 12-month post procedure evaluation. The follow-up visit assessment will include:

- Vital Signs (BMI, Blood Pressure, Heart Rate)
- NYHA Classification
- LAA Closure Imaging [CTA or TEE] \*
- Evaluation of AEs/SAEs
- Medications Review (Anticoagulants, antihypertensives, etc), including any adjustments

\*Prospective imaging (CTA/TEE) to be completed <u>at or after</u> the 12-month visit from the time of AtriClip implant. Retrospectively collected CTA or TEE may be submitted to the Core lab for review. Imaging that meets the quality of the Core Lab's acquisition protocol may be used in lieu of prospective imaging.

# 6.3.2 Study Exit

Once study subjects have completed their last follow-up visit, and TEE closure imaging has been obtained, the subject will be exited from the study.




# 6.3.3 Schedule of Events

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| Trial Activity | Baseline<br>(Within 30 days of index<br>procedure) | Index Procedure | 30-days Post-Procedure<br>(Within 23-37 days of<br>index procedure) | 12-months Post-Procedure<br>(≥ 12-months from index<br>procedure) |
| Informed Consent & Inclusion/Exclusion | х | | | |
| Demographics (Age, Sex, Race, Ethnicity) | X | | | |
| Vital Signs (BMI, BP, Heart Rate) | X | | | Х |
| Medical/Surgical/Cardiac History (CHADS, CHADSVASC, HASBLED scores) | х | | | |
| NYHA Classification | X | | х | Х |
| Intra-Op TEE, if done | | х | | |
| CTA or TEE Imaging | | | | Х |
| Cardiac Medications/Adjustment Review | x | | | Х |
| Adverse Events (AEs/SAEs) | | х | х | Х |
| Surgical Procedure | | х | | |

Note: Medications administered during the post-operative period do not need to be captured in the eCRF.




#### 6.4 Requirement for Clinical Laboratories

An independent Core Laboratory will be utilized for assessment LAA exclusion defined by the absence of residual communication (no leaks) and residual pocket (≤10 mm)) between the LA and LAA. Imaging for subjects include:

• CTA or TEE imaging at last follow-up visit (12-months or greater post-procedure visit)

All closure imaging submitted should be performed in accordance with the Core Laboratory's recommended protocol.

# 7 ADVERSE EVENTS

#### 7.1 Definition

#### 7.1.1 Adverse Event

Adverse Event (AE) is defined as any undesirable clinical occurrence or change from subject's baseline (or pre-device procedure) condition, whether it is considered device related or not. An AE is also defined by the International Organization for Standardization (ISO) as an untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated.

Adverse Event Identification: a condition that is one of the following:

- 1. A unique symptom or event that is a change from the subject's baseline status.
- 2. A series of symptoms or events that can be categorized as a single entity based on definitions found herein.
- 3. A specific diagnosis responsible for a clinical change.
- 4. A worsening or exacerbation of a pre-existing condition.

#### 7.1.2 Serious Adverse Event

If the AE meets any of the criteria below, it is regarded as a SAE.

- a) Led to a death,
- b) Led to a serious deterioration in health of the subject, that either resulted in
  - 1. Life-threatening illness or injury, or
  - 2. Hospitalization (initial or prolonged) or
  - 3. Disability or permanent impairment of a body structure or a body function
  - 4. Congenital anomaly (physical or mental)/birth defect/fetal distress/fetal death
  - 5. Chronic disease
  - 6. Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
- c) Other Serious (important Medical Events).

Events qualifying as SAEs as defined in section 4.1 include:

- Death
- Major bleeding (BARC 3 and above)
- Surgical site infection




- Pericardial effusion requiring intervention
- Clinical diagnosis of myocardial infarction

Any condition that was recorded as pre-existing is not a SAE unless there is a change in the nature, severity, or degree of the condition.

**Note:** A planned hospitalization for pre-existing condition, or a procedure required by the protocol, without a serious deterioration in health, is not considered to be an SAE.

Note: "Death" should not be reported as an adverse event. The cause of death should be reported as an adverse event. The only exception is "Sudden Death" when the cause is unknown.

## 7.1.3 Device Deficiency/Device Malfunction

Device Deficiency is defined as an inadequacy of a medical device related to its identity, quality, usability, durability, reliability, safety or performance, such as malfunction, misuse or use error and inadequate labeling. This includes the failure of the device to meet its performance specifications or otherwise perform as intended. Note: Performance specifications include all claims made in the labeling of the device.

A device malfunction is the failure of a device to meet its performance specifications or otherwise perform as intended.

All device deficiencies of the AtriClip LAA exclusion device shall be documented throughout the clinical investigation and managed by the sponsor in accordance with written procedures for the control of a non-conforming product. The sponsor shall take, where applicable, appropriate corrective and preventative actions to protect the safety of subjects, users, and other persons. Device deficiencies of the comparator, if applicable, shall be documented. Where applicable, the analysis of used or explanted investigational devices shall be included as supportive information.

#### 7.2 Pre-Existing Conditions Versus Adverse Events

A pre-existing condition is defined as a medical condition that is present before the index procedure and is to be reported as part of the subject's medical history. It must be reported as a new AE if the intensity, frequency, or the character of the condition worsens during the study treatment and the AE was determined to have the relationship to the study procedures and/or study devices.

To avoid confusing pre-existing conditions with AEs during data analysis, the study sites must make all attempts to provide start dates for all baseline medical conditions. Any pre-existing condition that now meets the stated criteria as an AE should be recorded on the AE CRF as an exacerbation of the pre-existing condition and the start date will be recorded as the time when the exacerbation occurred.

# 7.3 Severity of Adverse Events

It is the Investigator's responsibility to assess the severity of an AE. A change in severity may constitute a new reportable AE.




The following guideline should be used to determine the severity of each adverse event:

- MILD: Awareness of experience, but easily tolerated. No medical intervention required
- **MODERATE:** Enough discomfort to interfere with usual activities. Medical intervention required
- **SEVERE:** Inability to carry out usual activities. Medical/surgical intervention (including hospitalization or prolongation of hospitalization) required.

# 7.4 Device Relationship

Determination of whether there is a reasonable possibility that an investigational product or device under investigation caused or contributed to an AE is to be determined by the Investigator and recorded on the appropriate CRF form. Determination should be based on assessment of temporal relationships, evidence of alternative etiology, medical/biologic plausibility, and subject condition (pre-existing condition).

It is the Investigator's responsibility to assess the relationship of an AE to the study procedure and/or device.

Adverse events will be assigned an attribution according to the Investigator's believed primary cause. Events will be categorized by relationship to the investigational device(s) listed in this protocol or ancillary device, surgical ablation procedure, general cardiac surgical procedure or subsequent intervention, concomitant medications, pre-existing condition, intercurrent condition, intercurrent intervention, or unknown.

The following guidelines should be used in determining the relationship of an adverse event to the study device or procedure:

- **Unknown:** A clinical event (including abnormal laboratory result) that cannot be determined to be related or unrelated to device/procedure/drug given information provided.
- **Device Related Adverse Event**: An adverse event, that in the judgment of the Investigator, resulted from use or placement of the AtriCure AtriClip LAA Exclusion System and may have caused or contributed to the AE.
- Procedure Related Adverse Event: An adverse event which, in the judgment of the Investigator, results as a consequence of the procedure (surgical procedure or general cardiac surgical procedure, subsequent intervention) and is not specifically related to the use of the AtriCure AtriClip LAA Exclusion System.
- General Surgery Related Adverse Event: An adverse event which, in the judgement of the Investigator, results as a consequence of general cardiac surgical procedural complications and/or subsequent interventions.
- Concomitant Medication-Related Adverse Event: An adverse event is considered to be concomitant medication related when, in the judgment of the Investigator, it is reasonable to believe that the event is associated with concomitant medications used in conjunction with the AtriClip device and is not otherwise specific to the AtriClip device (e.g. bleeding associated with anticoagulation medication).
- **Intercurrent Condition**: It is reasonable to believe that the event is directly associated with an intercurrent condition/co-morbidity.




• **Intercurrent Intervention**: It is reasonable to believe that the event is directly associated with an intercurrent intervention which was performed for reasons other than to address a device or general cardiac surgical procedure related complication.

## 7.4.1 Unanticipated (Serious Adverse) Device Effect [U(S)ADE]

Unanticipated serious adverse device effect (USADE) refers to any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

# 7.5 Adverse Event and Device Deficiency/Device Malfunction Reporting

# 7.5.1 AE/ADE/UADE Reporting

## **General AE Reporting**

Safety surveillance and reporting starts as soon as the subject is enrolled in the clinical investigation. Safety surveillance and reporting will continue until the 12-Month follow-up visit has been performed, the subject is deceased, the subject concludes participation in the clinical investigation, or the subject withdraws from the clinical investigation. Except for those events listed in Section 7.6 all adverse event data potentially related to device or implant procedure, including deaths and device deficiency data, thromboembolic events, or events related to the 12-month TEE/CTA will be collected throughout the time period defined above and will be reported to the Sponsor on the eCRF. Additional information with regard to an adverse event should be updated within the appropriate CRF.

Standard medical terminology should be used when recording AEs.

In addition, the following information should be recorded:

- Onset Date
- Resolution date or date of death
- Intensity of the event
- Action Taken
- Outcome of the event
- Relationship of AE
- Indication of whether the event is serious

#### 7.5.2 SAE/USADE Reporting

The investigator (or designee) must report all SAE/USADEs to the Sponsor via the Adverse Event CRF as soon as possible but no later than outlined below.




| Clinical<br>Site | Reporting timelines |
|---|---|
| All Sites | SAEs must be reported to the Sponsor no later than 10 calendar days from the day the site personnel became aware of the event or as per the investigative site's local requirements, if the requirement is more stringent than those outlined. |
| | An event determined by the Investigator to be life-threatening or to have led to death must be reported within 24 hours. |

The date the site staff became aware the event met the criteria of an SAE must be recorded in the eCRF and ensure relevant source documents are collected. The Investigator will further report the SAE to the local IRB/EC according to the institution's IRB/EC reporting requirements. In the event of system outages or technical difficulties, serious and any unanticipated adverse events may be submitted via e-mail to <a href="mailto-sae-nail

The Investigator (or designee) shall send a written report including a narrative description of the serious and/or unanticipated adverse event to AtriCure or their designee within three (3) working days of the initial report. The Investigator should follow all unresolved serious adverse events until the events are resolved, or the subject has exited the study, or the adverse event is otherwise explained.

AtriCure, Inc., or their designee, in cooperation with the Investigator, will assess all serious adverse events considered device-related for potential report-ability to the FDA as an Unanticipated Adverse Device Effect (UADE) in accordance with 21 CFR Part 812.46(b).

If a UADE determination is made, the Investigator and Sponsor will comply with UADE reporting requirements per 21 CFR Part 812.150. The Sponsor shall report the results of such evaluation to FDA and to all reviewing IRBs/ECs and participating Investigators within thirty (30) working days after the Sponsor first receives notice of the UADE. Thereafter the Sponsor shall submit such additional reports concerning the effect as FDA requests. Similarly, the Investigator shall submit to their reviewing IRB a report of any UADE as soon as possible, but in no event later than ten (10) working days, (or per local IRB requirements) after the Investigator first learns of the effect. The Investigator (or designee) shall provide documentation of the UADE report/notification sent to their IRB to AtriCure (or designee).

Note: It is also the responsibility of the Investigator to inform their IRB of other SAEs (i.e. non-UADEs) as required by their IRB/EC procedures and in conformance with FDA requirements.

If the subject reports any device or procedure related adverse events that are potentially serious during the follow-up evaluation period, the subject should return to the investigator's facility for further evaluation of the event.

#### 7.5.3 Device Deficiency/Malfunction Reporting

All device deficiencies/malfunctions should be reported on the appropriate CRF.




The investigator should report all device deficiencies/malfunctions to the Sponsor as soon as possible but no later than outlined below.

| Clinical Sites | Reporting timelines |
|---|---|
| All Sites | Device deficiencies/malfunctions must be reported to the Sponsor no later than 10 calendar days from the day the site personnel became aware of the event or as per the investigative site's local requirements, if the requirement is more stringent than those outlined. |

# 7.5.4 Adverse Event Reporting to Country Regulatory Authorities by the Sponsor

The Sponsor will report SAEs and reportable device deficiencies/malfunctions to the country regulatory authority, per local requirements.

Clinical investigation SAEs and device deficiencies/malfunctions reportable per MedDEV 2.7/3 regulations will be submitted to European Competent Authorities by the Sponsor's Clinical Product Safety & Surveillance Group.

# 7.6 Expected Morbidity/Procedural Complications Reporting

For purposes of this study, the following events occurring within 48 hours of study procedures are not considered reportable (not recorded on eCRF but recorded in source documents) as they are normally expected to occur in conjunction with surgical treatment procedures or are associated with customary, standard care of subjects undergoing cardiac surgery:

- Chest pain without associated ECG changes
- Post-operative/post-procedure pain
- Post-anesthesia emesis, nausea, or headache (within 24 hours of procedure)
- Electrolyte imbalance without clinical sequelae following procedure, even if requiring correction
- Low grade temperature increase (101°F or 38.5°C)
- Dizziness: Imprecise term commonly used to describe various symptoms such as faintness, giddiness, imbalance, lightheadedness, unsteadiness or vertigo.
- Elevated white blood count, outside the standard laboratory normal value, without signs and symptoms of infection
- Post-operative hematocrit decreases from baseline measured in the OR, prior to the first incision, not associated with hemodynamic changes, remaining above 25% and requiring < 2 units PRBC's</li>
- Minor, localized tenderness, swelling, induration, oozing, etc. at surgical site.
- Sinus bradycardia/tachycardia that does not require treatment or intervention
- Systolic or diastolic blood pressure changes that do not require treatment or intervention.
- Any blood transfusions during preplanned operative procedures and unrelated to an adverse event.
- Thrombocytopenia: does not become an AE until treatment is administered.




- Atelectasis collapse of lung tissue affecting part or all of one lung; the alveoli are deflated. This is not considered to be an AE unless treatment other than chest PT is required or it prolongs hospitalization.
- Hyperglycemia The use of insulin in the post-operative period does not constitute
  hyperglycemia if during the same hospitalization. An elevated blood sugar of less than
  250 mg/dl during the first 48 hours post-operative does not constitute hyperglycemia.
- Pleural effusion is not an event unless treatment with thoracentesis or chest tube insertion is required
- Pericardial effusion without hemodynamic compromise or treatment
- Atrial Fibrillation /Atrial Flutter/Atrial Tachycardia with or without cardioversion.
- Junctional Rhythm requiring temporary pacing

Note: Treated subjects will have received general anesthesia and therefore will also be subject to general anesthesia-associated complications and morbidity. These are also not considered reportable (recorded on eCRF) adverse events.

Note: This listing of events is intended to provide guidance to the Investigator and investigational site for the purpose of adverse event reporting. The Investigator should utilize his/her own clinical judgment in evaluating adverse experiences and may decide that the above events should be reported as adverse events based on the IRB/EC reporting requirements or the subject clinical situation.

## 7.7 Product Complaints

A product complaint is any written electronic or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, usability safety, or performance of a device after it is release for distribution (a medical device that has been released from the organization's control or related to a service that affects the performance of such medical devices). Product complaints may or may not be associated with an AE.

# 7.7.1 Reporting Product Complaints

All product complaints (as defined above) related to an investigational product (shall be documented throughout the clinical investigation and appropriately managed by the sponsor. All reported device observations, malfunctions or failures for the AtriClip LAA Exclusion system are required to be documented in the EDC within 10 days of observation of the Product Complaint and sent via e-mail to <a href="mailto:pcomplaints@atricure.com">pcomplaints@atricure.com</a> by the PI or study staff.

If the AtriClip LAA Exclusion system or component is involved in a complaint, the device should be returned to AtriCure (e.g., product is damaged or use results in an AE). If this occurs, sponsor representatives will send a Used Product Return Kit to study site personnel for packaging the product; which (depending on the product) may be sent to the appropriate facility for decontamination and further investigation of the complaint.




# 7.7.2 Reporting Product Complaints with Non-Investigational Device Products

All reported device observations, malfunctions or failures for AtriCure Non-Investigational (i.e. Marketed Products) are required to be documented in the Clindex database on the device observation eCRF and emailed to <a href="mailto:pcomplaints@atricure.com">pcomplaints@atricure.com</a> within 10 days of the observation by the PI or study staff.

If an event involving an AtriCure device is subject to reporting under the Medical Device Reporting Regulation (MDR), AtriCure shall submit to the FDA the appropriate reports required by MDR within the timeframes identified in 21 CFR Part 803.

#### 7.7.3 Non-AtriCure Product Complaints

In compliance with the requirements of 21 CFR Part 803.30 (MDR), the study site (user facility) will be instructed to report any SAEs associated with the use of other (non-AtriCure) marketed products/devices in this study to the respective manufacturer and, if the SAE involves a death, the complaint should be reported to the manufacturer.

# 7.7.4 Reporting Product Complaints for Global Compliance

If a Product Complaint is reported in conjunction with a SAE/UADE, reporting guidelines will be the same as those listed in Section 7.5.4.

# 8 STATISTICAL CONSIDERATIONS

The following section describes the statistical methods for the clinical investigation. Additional details on statistical analyses, including justification of clinical investigation design, sensitivity analyses, pool-ability analyses, subgroup analyses etc., may be maintained in a separate Statistical Analysis Plan.

#### 8.1 Analysis Populations

# Intention-to-Treat Population:

The Intention-to-Treat (ITT) population consists of the subjects with AtriClip implant. This is the primary population for performance endpoints.

#### Protocol Population:

The Per-Protocol (PP) study population is defined by the ITT population but without any major protocol deviations, that is, those that could potentially bias the results. This population is defined for the primary performance endpoints.

#### 8.2 Statistical Analyses

The primary goal of the study is to demonstrate safety and performance of the Flex-V and PRO•V device. For the study to be successful, the safety and performance endpoints must be statistically significant relative to their respective performance goals.

Standard descriptive statistics will be used to summarize numeric variables, including the number of observed values, mean, standard deviation, median, minimum and maximum values.




Summaries of categorical variables will include the number and percentage of observed values, at each level of the categorical variable. Baseline and demographic information, including age, gender, race, ethnicity, BMI, and medical history will be summarized with standard descriptive statistics.

Two-sided 95% and 90% confidence intervals will be provided for point estimates as appropriate.

# 8.2.1 Primary Performance Endpoint Analysis

The primary performance endpoint is further defined in section 4.1 of the protocol.

Subjects meeting the primary performance endpoint (success LAA exclusion at least 12-months post AtriClip implant) will be labeled as "responders", and the proportion of responders will be compared to a performance goal (PG) of 80%.

An exact binomial test will be conducted at a one-sided  $\alpha$  = 0.025 level of significance to test the following hypothesis that the proportion of performance successes is significantly higher than the PG:

 $H_0: p \le 80\%$ 

 $H_A: p > 80\%$ 

where p is the responder rate at last follow-up visit occurring at least 12-months post-procedure. The ITT population will be the primary population for this analysis.

# 8.2.2 Primary Safety Endpoint Analysis

The primary safety endpoint is the proportion of subjects free from SAEs, as described in section 4.1 of the protocol, through 30-days post AtriClip implantation. The SAE rate will be compared against a PG of 10.5%.

An exact binomial test will be conducted at a one-sided  $\alpha = 0.05$  level of significance to test the following hypothesis that the proportion of MAEs is significantly lower than the PG:

The hypothesis test for the safety endpoint is:

 $H_0$ :  $q \ge 10.5\%$ 

 $H_A$ : q < 10.5%

where q is the proportion of subjects with MAEs through 30-days AtriClip implantation in the safety population. The ITT population will be the primary population for this analysis.

## 8.2.3 Secondary Endpoint Analyses

The secondary endpoints are described in section 4.3 of the protocol.

All analyses will be conducted using appropriate statistical methods as described in Section 8.2 and for the primary performance endpoint, as applicable. These will include analyses of the populations and subgroups as specified in this protocol and may also include additional endpoints, populations and/or subgroups.




# 8.2.4 Long-Term Safety Analyses

Serious events related to the index procedure (such as LAA tears, tissue injury or bleeding which requires intervention) will be reported. Descriptive statistics will be provided. No formal hypothesis testing will be done.

# 8.3 Sample Size Calculation and Assumptions

## **Performance Endpoint**

The 12-month LAA closure rate (No leak) for contemporary devices ranges from 66 % - 89.5%. (Kar, 2021) In-line with these rates, a PG of 80% is proposed for this study.

Based on the performance goal of 80% success and an expected success rate of 90%, a sample size of 143 subjects provides 92% power using a one-sided Exact test, with  $\alpha$  = 0.025 level of significance to demonstrate primary performance success. Assuming an attrition rate of 16% at the last follow-up visit post procedure, a total of 170 subjects will be enrolled.

The lowest primary performance endpoint that would meet the PG is 86.7% (that is, 124 out of 143 subjects are responders).

#### **Safety Endpoint**

Minimal to no missing data are expected for the primary safety. Based on a PG of 10.5%, and an expected population MAE rate of up to 5%, a sample size of 170 subjects will have 85.4% power using a one-sided Exact test, with at a one-sided  $\alpha$  = 0.05 level of significance.

The highest primary safety endpoint that would meet the PG would be 6.5% (that is, 11 out of 170 subjects experience at least one MAE).

Watchman FLX device is CE approved and improved safety when compared to previous iterations of this device (1) reported a safety rate of 5% (20/400) [95% one-sided upper confidence limit of 7%] reported within similar timeframe (45 days) after the device implant. The safety performance goal of 10.5% is based on 1.5 times the UCL of 7%.




## 8.4 Timing of Analysis

The primary performance endpoint analysis will be conducted when all subjects have completed at least their 12-months post-procedure visit. The expected duration of the study is approximately 21 months.

# 8.5 Subgroup Analysis

No subgroup analyses are planned for this clinical investigation. However primary safety and performance endpoints will be summarized by sex, race and other subgroups as needed.

#### 8.6 Multiplicity

No alpha multiplicity adjustments are planned for the exploratory and supporting secondary endpoints and analysis populations defined in the study.

#### 8.7 Pooling Strategy

For this study, data will be pooled from multiple study sites. The justification for pooling will be made on a clinical basis considering three factors: (1) the study sites must implement one common protocol, (2) the Sponsor must closely monitor study site compliance with the protocol, and (3) the study site must use common data collection procedures.

# 8.8 Procedures for Accounting for Missing Data

As applicable, several sensitivity analyses will be performed to evaluate the effect of the missing data on the primary performance and safety endpoints, including multiple imputation, last observation carried forward (LOCF) and a tipping point analysis. Details will be provided in the SAP prior to database lock.

## 8.9 Statistical Criteria for Termination

There are no statistical criteria for termination of this clinical investigation.

#### 8.10 Success Criteria

For the trial to be successful, the performance endpoints must be statistically significant relative to their respective performance goals and that the hypotheses are met. If the null effectiveness hypothesis is rejected, the treatment will be considered beneficial.

#### 8.11 Deviations from Statistical Plan

Any major changes to the statistical plan will be documented in an amendment to the statistical plan. Less significant changes to the planned analyses will be documented in the final report.

#### 9 <u>DIRECT ACCESS TO SOURCE DATA/DOCUMENTS</u>

The investigator/institution will permit direct access to source data/documents for the purpose of performing clinical investigation-related monitoring, audits, IRB/EC review and regulatory inspections.




Subjects providing Informed Consent are agreeing to allow clinical investigation monitors or regulatory authorities including foreign countries to review, in confidence, any records identifying the subjects in this clinical investigation. This information may be shared with regulatory agencies; however, Sponsor undertakes not to otherwise release the subject's personal and private information.

## 10 QUALITY CONTROL AND QUALITY ASSURANCE

# 10.1 Selection of Clinical Sites and Investigators

The Sponsor will select investigators qualified by training and experience to participate in the clinical investigation. Sites will be selected based upon review of a recent site assessment, if applicable, and the qualifications of the investigators who will participate in the clinical investigation.

## 10.2 Clinical Investigation Finances and Agreements

The clinical investigation will be financed by AtriCure. Investigational sites will be compensated by AtriCure for participation in the clinical investigation per the conditions of agreement between the Sponsor and the Investigational site.

#### 10.3 Protocol Amendments

Approved protocol amendments will be provided to the Investigators by the Sponsor prior to implementing the amendment. The Principal Investigator is responsible for notifying the IRB/EC or equivalent committee of the protocol amendment (administrative changes) or obtaining IRB's/EC's approval of the protocol amendment (changes in subject care or safety), according to the instructions provided by the Sponsor with the protocol amendment.

Acknowledgement/approval by the IRB/EC of the protocol amendment must be documented in writing prior to implementation of the protocol amendment. Copies of this documentation must also be provided to the Sponsor.

The protocol and all subsequent amendments to the protocol are prepared by the Sponsor, agreed upon between the Sponsor and the National Principal Investigator, accepted by all Principal investigators, and are recorded with a justification for each amendment.

#### 10.4 Training

#### 10.4.1 Site Training

All Investigators and clinical investigation personnel are required to attend Sponsor training sessions, which may be conducted at an Investigator's meeting, an onsite initiation visit, a virtual site initiation visit or other appropriate training sessions. Over-the-phone or self-training may take place as required. Training of Investigators and clinical investigation personnel will include, but is not limited to, the protocol requirements, investigational device usage, electronic case report form completion and clinical investigation personnel responsibilities.




All Investigators and clinical investigation personnel that are trained must sign a training log (or an equivalent) upon completion of the training. Prior to signing the training log, Investigators and clinical investigation personnel must not perform any protocol-related activities that are not considered standard of care at the site.

## 10.5 Monitoring

Sponsor and/or designee will monitor the clinical investigation over its duration according to the protocol specific monitoring plan which will include the planned extent of source data verification.

Prior to initiating any procedure, the Sponsor monitor (or delegate) will ensure that the following criteria are met:

- The Investigator understands and accepts the obligation to conduct the clinical investigation according to the protocol and applicable regulations, and has signed Clinical Study Agreement
- Source documentation (including original medical records) must be available to substantiate proper Informed Consent procedures, adherence to protocol procedures, adequate reporting and follow-up of adverse events, accuracy of data collected on case report forms, and device information.
- The Investigator/site will permit access to such records. A monitoring visit sign-in log will be maintained at the site. The Investigator will agree to dedicate an adequate amount of time to the monitoring process. The Investigator and/or research coordinator will be available for monitoring visits. It is expected that the Investigator will provide the monitor with a suitable working environment for review of clinical investigation-related documents.

This study will be monitored by the sponsor to ensure:

- The rights and well-being of the subjects are protected;
- The reported study data is accurate, complete, and verifiable from source documents;
- The conduct of the study is in compliance with the currently approved protocol and amendment(s), applicable GCPs, and with applicable local and regional regulatory requirements.

#### 10.6 Protocol Deviations

Protocol deviations are events occurring during the conduct of the study which are not in compliance with the protocol and for which an amendment has not been granted. The Investigator should not deviate from the protocol for any reason except in cases of medical emergencies when the deviation is necessary to protect the rights, safety and well-being of the subject or eliminate an apparent immediate hazard to the subject. In that event, the Investigator will notify Sponsor immediately by phone or in writing.

For retrospective data collection, it is possible that subject visits post-procedure will vary based on institutional standard of care. For the purposes of this study individual protocol deviation waivers will not be required for the following:

• any retrospective subject visit that falls outside of the protocol defined visit window will not be documented as a protocol deviation; and



• Vital signs, Intra-Op TEE, or NYHA classifications that were not retrospectively performed will not be documented as a protocol deviation.

All deviations must be reported to the Sponsor using the Deviation CRF. The occurrence of protocol deviations will be monitored by the Sponsor for evaluation of investigator compliance to the protocol and regulatory requirements and dealt with according to written procedures. Investigators will inform their IRB/EC or equivalent committee of all protocol deviations in accordance with their specific IRB/EC or equivalent committee reporting policies and procedures.

In the event of repeated non-compliance, as determined by the Sponsor, a Sponsor's monitor or company representative will attempt to secure compliance by one or more of the following (and not limited to):

- Visiting the Investigator and/or delegate
- Telephoning the Investigator and/or delegate
- Corresponding with the Investigator and/or delegate

Repeated non-compliance with the signed agreement, the protocol or any other conditions of the clinical investigation may result in further escalation in accordance with the Sponsor's written procedures, including securing compliance or, at its sole discretion, Sponsor may terminate the Investigator's participation in the clinical investigation.

# 10.7 Quality Assurance Audit

A Sponsor representative or designee may request access to all clinical investigation records, including source documentation, for inspection during a Quality Assurance audit.

In the event that an Investigator is contacted by a Regulatory Agency in relation to this clinical investigation, the Investigator will notify Sponsor immediately. The Investigator and Research Coordinator must be available to respond to reasonable requests and audit queries made during the audit process. The Investigator must provide Sponsor with copies of all correspondence that may affect the review of the current clinical investigation (e.g., Form FDA 483, Inspectional Observations, Warning Letters, Inspection Reports, etc.). The Sponsor may provide any needed assistance in responding to regulatory audits.

### 10.8 Committees

The Sponsor shall ensure oversight of any clinical investigation-related duties and functions. The outsourcing of duties or functions to external organizations, including subcontractors of the Sponsor's CRO(s)/Committees, shall be addressed by the Sponsor in accordance with written procedures for control of suppliers and/or charters as applicable. Additionally, records of transfer of duties and functions shall be maintained where applicable.

#### 10.8.1 Study Oversight Committee

The Study Oversight Committee is comprised of the National PI and Sponsor Medical Advisor. The Chairman of the Core laboratories and other Sponsor personnel may also participate in the




Committee meetings if appropriate. Meeting minutes from this committee will be filed with the sponsor.

The Study Oversight Committee is responsible for overseeing the scientific and operational aspects of the clinical investigation.

Specifically, the committee with participate and/or advise on the following:

- Review of the study protocol
- Review of the training material for the sites as applicable
- Study operations and safety
- Discussion of study related issues with the sites, as needed
- Regulatory communication, as needed

#### **10.8.2 Publications Committee**

A Publication Committee may be established to oversee clinical investigations publications, including publication planning and authorship determinations. Publication Committee membership may include the National PI(s), Site Principal Investigators, a representative of the Sponsor and a statistician. The Publication Committee will determine policy and strategies regarding individual presentations and/or publications arising from clinical investigation generated data. The committee will also review all external requests for accessing clinical investigation-related data and strategies aligning with the Sponsor's presentation and publication team expectations.

# 10.8.3 Independent Physician Adjudicator (IPA)

An independent, non-investigator physician(s) will function as the adjudicator(s) under the direction of AtriCure, Inc. The physician(s) will be responsible for the review and adjudication of the following:

- 1. All Serious Adverse Events listed under the primary endpoint;
- 2. All Unanticipated Device Effects:
- 3. All Adverse Events that are potentially related to the procedure or any of the AtriCure AtriClip devices used in the study;

In addition, all primary endpoints and other adverse events determined by the adjudicator(s) to be relevant, will be adjudicated until the subject exits the study.

#### 11 DATA HANDLING AND RECORD KEEPING

The Sponsor and/or its affiliates will maintain documentation of the systems and procedures used in data collection for the duration of the clinical investigation.

CRF data collection will be performed through a secure web portal and only authorized personnel will access the Electronic Data Capture (EDC) system using a unique username and password to enter, review or correct data. Passwords and electronic signatures will be strictly confidential.




The data will be subjected to consistency and validation checks within the EDC system and supplemental review by the Sponsor.

At the conclusion of the clinical investigation, completed CRF images with the date-and-time stamped electronic audit trail indicating the user, the data entered, and any reason for change (if applicable) will be provided to the investigational sites.

For the duration of the clinical investigation, the Investigator will maintain complete and accurate documentation including, but not limited to, medical records, clinical investigation progress records, laboratory reports, CRFs, signed ICFs, correspondence with the IRB/EC and clinical investigation monitor/Sponsor, adverse event reports, and information regarding subject discontinuation or completion of the clinical investigation.

The Investigator shall assure the accuracy, completeness, legibility and timelines of the data reported to the sponsor on the CRFs and in all required reports. All copies of the retained original source documents shall be certified, as indicated by a dated signature by a member of the investigation site team unless generated through a validated process.

# 11.1 Protection of Personally Identifiable Information

The Sponsor respects and protects personally identifiable information collected or maintained for this clinical investigation.

The Sponsor implements technical and physical access controls to ensure that Personal Information is accessible only to and processed only on a 'need to know' basis, including periodic review of access rights, and revocation of access when an individual's employment is terminated or the individual transitions to a role that does not require access to Personal Information, and appropriate restrictions on physical access to premises, facilities, equipment, and records containing Personal Information.

The Sponsor requires the investigational sites to transfer into Sponsor's data management systems only pseudonymous Personal Information necessary to conduct the Clinical Investigation, such as the subject's medical condition, treatment, dates of treatment, etc. The Sponsor discloses as part of the clinical investigation Informed Consent process that some Sponsor representatives still may see Personal Information at the participating sites for technical support of the participating physicians on the procedures, monitoring and quality control purposes. Confidentiality of Personal Information will be observed by all parties involved at all times throughout the clinical investigation. The privacy of each subject and confidentiality of his/her information will be preserved in reports and when publishing any data.

The Sponsor data management systems and processes were designed, developed, and tested according to industry standards to appropriately safeguard Confidential Information (including any Personal Information) against unauthorized access and/or interference by third parties, intrusion, theft, destruction, loss or alteration. Clinical Investigation data are encrypted in transit and at rest.




#### 11.2 Data Management Plan

A Data Management Plan (DMP) will describe procedures used for data review, data cleaning, and issuing and resolving data discrepancies. If appropriate, the DMP may be updated throughout the duration of the clinical investigation. All revisions will be tracked and document controlled.

#### 11.3 Source Documentation

Regulations and GCP require the Investigator to maintain information in the subject's original medical records that corroborates data collected on the CRFs. In order to comply with these regulatory requirements/GCP, the following information should be included in the subject record at a minimum and if applicable to the clinical investigation:

- Medical history/physical condition of the subject before involvement in the clinical investigation sufficient to verify protocol entry criteria
- Dated and signed notes on the day of entry into the clinical investigation referencing the Sponsor, protocol number, subject ID number and a statement that Informed Consent was obtained
- Dated and signed notes from each subject visit (for specific results of procedures and exams)
- Adverse events reported and their resolution, including supporting documents, such as discharge summaries, catheterization laboratory reports, ECGs, and lab results including documentation of site awareness of SAEs and of investigator assessment of device relationship for SAEs.

#### 11.4 Case Report Form Completion

Primary data collection based on source-documented hospital and/or clinic chart reviews will be performed clearly and accurately by site personnel trained on the protocol and CRF completion. The investigator will ensure accuracy, completeness, legibility and timeliness of the data reported to the Sponsor on the CRFs and in all required reports.

CRF completion guidelines may also be developed to provide instructions to the site for accurate completion, correction and signature of CRFs along with expectations on handling clinical investigation deviations and unknown data, thus reducing the need of sponsor data queries. Only authorized site personnel will be permitted to enter the CRF data through the EDC system deployed by the Sponsor. An electronic audit trail will be used to track any subsequent changes of the entered data.

#### 11.5 Record Retention

The Sponsor and Investigator/Site will archive and retain all documents pertaining to the clinical investigation as per the applicable regulatory record retention requirements.

If custody of the records is transferred, notice of such a transfer should be given to the Sponsor no later than ten (10) working days after the transfer occurs.

The Investigator should retain copies of all documents pertaining to this clinical investigation (including source documentation, the Informed Consent document, and any other documents to




identify the subjects) for at least 2 years after this clinical investigation is completed. In addition, if the Clinical Investigator moves/retires, etc., he/she should provide AtriCure Inc. the name and address of the person who will look after and be responsible for the subjects' clinical investigation related records.

# 11.6 Investigational Devices Accountability

Subjects enrolled in this study will already have been treated, therefore device accountability is not required.

#### 12 ETHICAL CONSIDERATION

# 12.1 Institutional Review Board/Medical Ethics Committee Review and Approval

Institutional Review Board (IRB)/ Ethics Committee (EC) approval for the protocol and ICF/other written information provided to the subject will be obtained by the Principal Investigator at each investigational site prior to consenting and enrolling subjects in this clinical investigation. The approval letter must be received prior to the start of this clinical investigation and a copy must be provided to the Sponsor.

The IRB/EC may require a draft of the Clinical Study Agreement and proposed compensation to the investigation site or Principal Investigator be provided, including a letter of the Sponsor confirming outsourcing of duties and functions and CVs of the investigational site team.

Any amendments to the protocol as well as associated ICF changes will be submitted to the IRB/EC and written approval obtained prior to implementation, according to each institution's IRB/EC requirements.

No changes will be made to the protocol or ICF or other written information provided to the subject without appropriate approvals, including IRB/EC, the Sponsor, and the regulatory agencies (if applicable).

Until the clinical investigation is completed, the Investigator will advise his/her IRB/EC of the progress of this clinical investigation, per IRB/EC requirements. Written approval must be obtained from the IRB/EC yearly to continue the clinical investigation, or according to each institution's IRB/EC requirements.

No investigative procedures other than those defined in this protocol will be undertaken on the enrolled subjects without the written agreement of the IRB/EC and the Sponsor.

In accordance with the Declaration of Helsinki, a description of the clinical investigation shall be registered in a publicly accessible database before the start of recruitment activities and the content shall be updated throughout the conduct of the clinical investigation and the results entered at completion of the clinical investigation. Note: National regulations can apply concerning the timing of registration or updating the contents.




#### 13 CLINICAL INVESTIGATION CONCLUSION

The clinical investigation will be concluded when:

- All sites are closed AND
- The final report has been provided to investigators or the Sponsor has provided formal documentation of clinical investigation closure.

# 14 PUBLICATION POLICY

The data and results from the clinical investigation are the sole property of the Sponsor. The Sponsor shall have the right to access and use all data and results generated during the clinical investigation. The Investigators will not use this clinical investigation-related data without the written consent of the Sponsor for any purpose other than for clinical investigation completion or for generation of publication materials, as referenced in the Clinical Study Agreement. Single-center results are not allowed to be published or presented before the multi-center results. Any proposals for publications or presentations by the investigators must be reviewed and approved by the Sponsor in a timely manner to enable Sponsor review in compliance with the Sponsor's publication policy set forth in the Clinical Study Agreement.

The Sponsor will be responsible for determining whether to register the clinical investigation on www.clinicaltrials.gov or any other clinical trials, in accordance with the International Committee of Medical Journal Editors guidelines, or any other applicable guidelines. In the event Sponsor determines that the clinical investigation should be registered, Sponsor shall be responsible for any such registration and results posting as required by the ClinicalTrials.gov website. Institution and/or Principal Investigator(s) shall not take any action to register the clinical investigation.

#### 15 RISK ANALYSIS

Surgical cardiac procedures are commonly performed and LAA exclusion is a well-accepted treatment, with a well-established risk profile. The primary objective of this study is to evaluate the long-term performance and safety of the AtriClip FLEX-V and PRO•V LAA Exclusion devices for exclusion of the left atrial appendage.

#### 15.1 Anticipated Clinical Benefits

The potential benefit to study subjects outweighs the risks of participation in this study. The benefits may include but are not limited to, the following:

• Overall advancement of medical and scientific knowledge that may benefit future subjects with similar conditions may be gained through this clinical study.

There may also be other benefits that are unforeseen at this time.

#### 15.2 Foreseeable Adverse Events and Anticipated Adverse Device Effects

Complications that could specifically have occurred at any time during the procedure, post procedure or may be possible during the follow-up period with the AtriCure AtriClip LAA Exclusion System. Refer to Appendix IV for a listing of foreseeable adverse events.




# 15.3 Residual Risks Associated with the Device Under Investigation, as Identified in the Risk/Quality Management Report

Subjects enrolled in this trial have already been treated, however risk analyses and evaluations of the device hazards and product design, application, and process have been conducted for the AtriClip LAA Exclusion System devices.

Upon review of the risk documentation for the AtriClip LAA Exclusion System, all individual residual risks were controlled and reduced to as far as possible. An acceptable level per the risk acceptability criteria set forth in the risk management plan was achieved.

#### 15.4 Risks Associated with Participation in this Clinical Investigation

The clinical investigation has been designed to involve as little pain, discomfort, fear, and any other foreseeable risk as possible for subjects.

# 15.5 Steps Taken to Control or Mitigate Risks

In-depth recommendations and special precautions are included in the IFU. Risks associated with this clinical investigation are minimized through investigator selection and training, prespecified subject eligibility requirements, and study monitoring to ensure adherence to the protocol. All adverse events and device deficiencies will be reported to the Sponsor and will be monitored internally for safety surveillance purposes.

#### 15.6 Risk to Benefit Rationale

The cumulative effect of all residual risks have been evaluated to ensure the overall residual risk of the product is acceptable and that the benefits of the device outweigh the overall residual risk.




# **APPENDIX I: REFERENCES**

- 1. Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, et al. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J 2012;33:2719–47. doi:10.1093/eurhearti/ehs253
- 2. Ailawadi, Gorav et al. "Exclusion of the left atrial appendage with a novel device: early results of a multicenter trial." *The Journal of thoracic and cardiovascular surgery* vol. 142,5 (2011): 1002-9, 1009.e1. doi:10.1016/j.jtcvs.2011.07.052
- 3. Calkins, Hugh et al. "HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for personnel, policy, procedures and follow-up. A report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation developed in partnership with the European Heart Rhythm Association (EHRA) and the European Cardiac Arrhythmia Society (ECAS); in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), and the Society of Thoracic Surgeons (STS). Endorsed and approved by the governing bodies of the American College of Cardiology, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, and the Heart Rhythm Society." Europace: European pacing, arrhythmias, and cardiac electrophysiology: journal of the working groups on cardiac pacing, arrhythmias, and cardiac cellular electrophysiology of the European Society of Cardiology vol. 9.6 (2007): 335-79. doi:10.1093/europace/eum120
- 4. Caliskan, Etem et al. "Epicardial left atrial appendage AtriClip occlusion reduces the incidence of stroke in patients with atrial fibrillation undergoing cardiac surgery." Europace: European pacing, arrhythmias, and cardiac electrophysiology: journal of the working groups on cardiac pacing, arrhythmias, and cardiac cellular electrophysiology of the European Society of Cardiology vol. 20,7 (2018): e105-e114. doi:10.1093/europace/eux211
- **5.** Ueberham, Laura et al. "Pharmacological and Non-pharmacological Treatments for Stroke Prevention in Patients with Atrial Fibrillation." *Advances in therapy* vol. 34,10 (2017): 2274-2294. doi:10.1007/s12325-017-0616-6
- **6.** van Laar, Charlotte et al. "Thoracoscopic Left Atrial Appendage Clipping: A Multicenter Cohort Analysis." *JACC. Clinical electrophysiology* vol. 4,7 (2018): 893-901. doi:10.1016/j.jacep.2018.03.009
- **7.** Healey, Jeff S et al. "Left Atrial Appendage Occlusion Study (LAAOS): results of a randomized controlled pilot study of left atrial appendage occlusion during coronary bypass surgery in patients at risk for stroke." *American heart journal* vol. 150,2 (2005): 288-93. doi:10.1016/j.ahj.2004.09.054
- 8. Kar et al. Primary outcomes evaluation of a next-generation left atrial appendage closure device. Results form PINNACLE FLX Trial. Circulation Volume 143, Issue 18, 4 May 2021; Pages 1754-1762




# **APPENDIX II: ABBREVIATIONS AND ACRONYMNS**

| Acronyms/Abbreviation | i erms |
|-----------------------|--------|
| • | |

AAD Antiarrhythmic Drug

ACC American College of Cardiology

ACT Activated Clotting Time
ADE Adverse Device Effect

AE Adverse Event

AEF Atrio-esophageal Fistula
AHA American Heart Association
ANC Absolute Neutrophil Count

ARDS Acute Respiratory Distress Syndrome

AV Atrioventricular

AVNRT Atrioventricular Nodal Reentry Tachycardia
BARC Bleeding Academic Research Consortium

BMI Body Mass Index

CEC Clinical Events Committee
CFR Code of Federal Regulations
CABG Coronary Artery Bypass Graft
CTA Computed Tomography Angiogram

CVA Cerebrovascular Accident

DCCV
DC Cardioversion
DOE
Dyspnea on Exertion
DVT
Deep Vein Thrombosis
ECG
Electrocrdiography
EDC
Electronic Data Capture
eCRF
Electronic Case Report Form

ECAS European Cardiac Arrythmia Society

EC Ethics Committee

EHRA European Heart Rhythm Association

EP Electrophysiology

ESC European Society of Cardiology FDA Food and Drug Administration

GCP Good Clinical Practice
GFL Glomerular filtration rate

GI Gastrointestinal HCT Hematocrit

HIPAA Health Insurance Portability and Accountability Act

HIT Heparin Induced Thrombocytopenia

HRS Heart Rhythm Society

ICD Implantable cardioverter-defibrillator

ICF Informed Consent Form




ICH International Conference on Harmonization

IDEInvestigational Device ExemptionILRImplantable Loop RecorderINRInternational Normalized RatioIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent to Treat LA Left atrium

LAA Left Atrial Appendage

LVEF Left Ventricular Ejection Fraction

MAE Major Adverse Event
MDR Medical Device Reporting
MI Myocardial Infarction
OAC Oral Anticoagulant
PE Pulmonary Embolism
PI Principal Investigator

PP Per Protocol

PHI Personal Health Information Permanent Pacemaker PPM **PRBC** Packed Red Blood Cells SAE Serious Adverse Event SAP Statistical Analysis Plan **SMP** Safety Monitoring Plan Shortness of Breath SOB Standard of Care SOC

TEE Transesophageal Echocardiogram (graphy)

TIA Transient Ischemic Attack

TTE Transthoracic Echocardiogram (graphy)
UADE Unanticipated Adverse Device Effect

ULN Upper Limit of Normal

USADE Unanticipated Serious Adverse Device Effect




# **APPENDIX III: DEFINITIONS**

# **BLOOD AND LYMPHATIC SYSTEM DISORDERS**

**Severe anemia**: Hematocrit below 25%. Generally, an accepted value to consider the need for transfusion of red blood cells. This is not in the setting of acute persistent bleeding.

Coagulopathy: Bleeding in the presence with abnormal clotting studies.

**Hemodilutional Anemia**: Anemia associated with fluid volume overload as a result of cardiopulmonary bypass.

**HIT (Heparin Induced Thrombocytopenia):** Low blood platelet count as a result of the medication heparin. Must have lab evidence of HIT +.

**Leukopenia:** Leukopenia is defined as leukocyte count of < 3.5 x10<sup>9</sup>/liter for more than 3 days.

**Neutropenia:** Neutropenia is defined as ANC <1000 per mm<sup>3</sup> for more than 3 days.

**Thrombocytopenia:** A persistent decrease in the number of blood platelets. This is not considered to be an AE until treated.

# **CARDIAC DISORDERS**

#### **Arrhythmias**

**Bradycardia**: Abnormally low heart rate (<60 bpm) requiring treatment (implantation of a temporary or permanent pacemaker, or medication).

**SVT:** Tachycardia in which QRS is narrow and P waves are present and associated. In certain SVT's the QRS may be wide (>120msec) when it is aberrant and in some the P wave may be invisible as it maybe superimposed on the QRS (AV Nodal Reentrant Tachycardia).

**Ventricular tachycardia (VT)**: A regular heart rhythm originating from the ventricle with a heart rate of greater than 100 bpm for at least 30 seconds or requiring termination due to hemodynamic compromise.

**Ventricular fibrillation (VF):** A rapid irregular ventricular rhythm due to multiple reentrant activities associated with essentially zero cardiac output.

#### Atrioventricular (AV) Block:

2<sup>nd</sup> degree: Second-degree (AV) block is characterized by interruption of impulse




conduction through the AV node. This may take the form of progressive prolongation of the P-R interval until there is a non-conducted beat with no QRS (Mobitz I or Wenckebach) or intermittent non-conducted P waves without preceding prolongation of the P-R interval or subsequent shortening of the interval (Mobitz II). This excludes block due to premature atrial beats

• **3**<sup>rd</sup> **degree**: Third-degree AV block (complete heart block) exists when more P waves than the QRS complexes exist and no relationship exists between them (no conduction).

**Angina**: A tight or heavy feeling in the chest, discomfort which spreads from the chest to the arm, back, neck, jaw, or stomach, numbness or tingling in the shoulders, arms or wrists, shortness of breath, and nausea.

Atrial thrombus: Thrombus formation or detection within the atrium.

**Cardiac Arrest:** Absent or inadequate contraction of the left ventricle of the heart that immediately causes body wide circulatory failure.

Cardiac Tamponade: See Cardiac Tamponade/Perforation definition.

Cardiac Tamponade/Perforation: Cardiac tamponade/perforation is defined as a complication of AF ablation if the development of a significant pericardial effusion occurs during or within 30 days of undergoing an AF Ablation procedure. A significant pericardial effusion is one which results in hemodynamic compromise, requires elective or urgent pericardiocentesis, or results in a pericardial effusion of 1 cm or more (by echocardiography). Cardiac tamponade/perforation should be classified as "early" or "late" depending on whether it is diagnosed during or following initial discharge from the hospital.

**Cardiogenic Shock**: Subject exhibits cardiogenic shock (systolic pressure < 80mm Hg and PCWP > 20mm Hg or cardiac index <1.8 liters/minute/m<sup>2</sup> or intra-aortic balloon pump or intravenous inotropes are needed to maintain a systolic pressure>80 mm Hg) for any time within 24 hours prior to index procedure.

**Congestive Heart Failure:** Documentation of one of the following:

- Paroxysmal nocturnal dyspnea (PND)
- Dyspnea on exertion (DOE) due to heart failure
- Elevated PCW with associated SOB or x-ray consistent with congestion.
- May be related to fluid overload in the presence of underlying cardiovascular disease.

**Heart Failure:** A clinical syndrome resulting from a cardiac disease which comprises ventricular systolic or diastolic function or both. Heart failure results when the heart is unable to generate a cardiac output sufficient to meet the demands of the body without unduly increasing diastolic pressure. Heart failure may be manifested by symptoms of poor tissue perfusion alone (i.e., fatigue, poor exercise tolerance, confusion) or by both symptoms of poor tissue perfusion and




congestion of vascular beds (e.g., dyspnea, chest rales, pleural effusion, pulmonary edema, distended neck veins, congested liver, peripheral edema). We will not distinguish between congestive and chronic heart failure for purposes of this protocol.

**Myocardial Infarction in the context of surgical AF Ablation**: The presence of any one of the following criteria:

- 1. Detection of ECG changes indicative of new ischemia (new ST-T changes), which may persist for more than one hour;
- 2. Development of new pathological Q waves on an ECG;
- 3. Imaging evidence of new loss of viable myocardium or new regional wall abnormality.

**Myocardial Perforation**: See Cardiac Tamponade/Perforation definition.

**Pericardial effusion**: Fluid detected in the pericardial space by standard imaging techniques (e.g., echocardiography).

**Pericarditis**: Irritation or inflammation of the pericardium associated with pain on inspiration and shortness of breath. Clinical signs may include shallow respiration, pericardial friction rub and ECG changes (ST elevation across the precordial leads).

**Sick sinus syndrome**: also called sinus node dysfunction, is a group of abnormal heart rhythms (arrhythmia) presumably caused by a malfunction of the sinus node, the heart's primary pacemaker.

**Unstable Angina**: Angina which increases in frequency, intensity, or duration, which occurs at rest, or which is new in onset. Unstable angina is a syndrome that is intermediate between stable angina and myocardial infarction: it is characterized by an accelerating or "crescendo" pattern of chest pain that lasts longer than instable angina, occurs at rest or with less exertion than instable angina, or is less responsive to medication. Unstable angina and myocardial infarction are considered acute coronary syndromes.

#### GASTROINTESTINAL/GENITOURINARY DEFINITIONS

**Atrioesophageal Fistula**: A connection between the atrium and the lumen of the esophagus. Evidence supporting this diagnosis includes documentation of esophageal erosion combined with evidence of a fistulous connection to the atrium such as an air embolus, an embolic event, or direct observation at the time of surgical repair. A CT scan or MRI scan are the most common methods of documentation of an atrial esophageal fistula. Esophagoscopy should NOT be performed as it may result in air insufflation into the left Atrium.

**Aortoesophageal Fistula**: Abnormal passage from aorta communicating with the esophagus (for the purposes of the protocol - likely resulting from an esophageal perforation or burn). Presentation of aortoesophageal fistula may include hematemesis (possibly massive). Diagnosis




may be obtained with a contrast CT scan, aortography, esophagoscopy, or barium swallow. A possible outcome of aortoesophageal fistula is sepsis, which may be diagnosed with blood cultures.

**Esophageal Dyskinesia**: diffuse spasms of the esophagus which may occur as the result of vagal nerve injury

**Esophageal Injury**: Any evidence of a mild complication such as erosion or ulceration or a major complication such as puncture, dissection, or perforation to the esophagus.

**Hernia**: an anatomical part (such as section of the intestine) protrudes through an opening, tear, or weakness in the abdominal wall musculature.

**Gastric Motility Disorders**: multiple gastric disorders may occur post AF ablation such as constipation, atony, weight loss, early satiety, diarrhea or GI disturbance.

**Gastroparesis:** delayed gastric emptying resulting in paresis of the stomach. As the vagus nerve controls the contractions of the stomach, this may occur when the vagus nerve is damaged and the muscles of the stomach and intestines do not work normally.

# **Renal Complications:**

- **Renal Failure:** Inability of the kidneys to filter toxins resulting in a serum creatinine increase to > 2.0 mg/dl and one of the following:
  - o increase of 2.0 mg/dl in serum creatinine over any previous value
  - $_{\odot}~$  50% or greater increase in creatinine over baseline procedural value requirement for dialysis
- Renal failure that requires dialysis: a significant decrease in renal function requiring dialysis.
- Renal Insufficiency: An increase in serum creatinine of ≥1.0 mg/dl over previous value.

**Vomiting:** The ejection of matter from the stomach in retrograde fashion through the esophagus and mouth.

# **GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS**

**Atypical Chest Pain**: Located under the sternum, left chest, abdomen, back, or arm and is fleeting or sharp. It is unrelated to exercise, not relieved by rest or the administration of nitroglycerin.

**Drug Reactions:** An unwanted or harmful side effect experienced following the administration of a drug or combination of drugs and is suspected to be related to the drug.




**Fatigue/Malaise:** Weariness, tiredness, or lack of energy. Generalized feeling of discomfort, illness, or lack of well-being.

**Fever:** A temperature > 101°F not related to a culture positive infection.

**General Discomfort**: Physical or psychosocial signs or symptoms commonly associated with hospitalization that are investigated and determined to require minor (i.e., aspirin, non-narcotic medication) or no treatment.

**Medication** Reaction: An unwanted or harmful side effect experienced following the administration of drug or combination of drugs and is suspected to be related to the drug.

**Multi-organ failure:** Failure of more than one organ due to shock or sepsis. This requires volume and inotropic support and has a high incidence of death.

Nausea: The unsettling feeling in the stomach that accompanies the urge to vomit.

**Non-ischemic Chest Pain:** Any discomfort in the chest, shoulder, back or chest wall for which a cardiac ischemic origin is ruled out or not suspected. May be cardiac (for example pericardial) or non-cardiac (for example gastrointestinal) in origin.

**Pain:** Reports of pain, ranging from mild discomfort to acute agony, may be generalized or localized, requiring treatment or intervention.

**Peripheral Edema**: is the swelling of tissues, usually in the lower limbs, due the accumulation of fluids.

**Reoperation:** A repeat operation for the same condition in the same subject or to resolve an adverse event resulting from the initial operation. Reoperation is not an adverse event – it is an outcome – the reason for reoperation is the adverse event.

**Sudden Death**: Cardiac arrest which is unexpected and occurs within minutes of the onset of symptoms.

**Death**: All-cause mortality. Death is not an adverse event, it is an outcome. The Adverse Event is what caused the death.

#### **HEPATOBILIARY DISORDERS**

**Hepatic Failure**: A clinical condition that results from severe and extensive damage of liver cells leading to failure of the liver to function normally and can induce mental confusion of various




degrees. Liver failure is described as the combination of hyperbilirubinemia (total Bilirubin > 2), coagulopathy with INR level greater than the upper limits of normal (in the absence of Warfarin (Coumadin) treatment) and hypoalbuminemia (Albumin < 3).

# **IMMUNE SYSTEM DISORDERS**

**Allergic Reaction**: A reaction to a foreign protein characterized by rash, nausea, vomiting, upper respiratory congestion, urticaria, shortness-of-breath, or general collapse (anaphylaxis).

# INFECTIOUS/INFLAMMATORY DEFINITIONS

**Bacteremia:** Presence of viable bacteria in the circulating blood without systemic manifestation (sepsis).

**Endocarditis**: An infection for which no source is identified associated with classic signs of endocarditis (positive blood cultures, fever, red blood cell casts in urine, splinter hemorrhages in finger nails, roof of mouth, lesions on retina, etc.) associated with a vegetation inside the atrium or on a valve which may be confirmed in echocardiography.

**Infection:** The following are the categories for infections:

- Deep Sternal: involving muscle, bone, and/or mediastinum
- **Deep Sternal Wound Infection**: Infection involving the sternum and/or mediastinum as documented by clinical examination and culture which may require reoperation with sternal debridement and/or sternal rewiring.
- Lung: involving airways associated with intubation or other respiratory causes
- Leg: involving a leg vein harvest site.
- **Major:** Including the chest wall, heart valves, mediastinum, etc., culture proven infection or presumptive treatment with antibiotics for clinically diagnosed infection
- **Minor:** Temperature > 101°F /38.5°C or higher and a positive culture (e.g., tissue, urine, etc.)
- Or Systemic Infection: Bloodstream infection caused by bacteria.

**Mediastinitis**: The diagnosis requires at least one of the following: (1) an organism isolated from culture of mediastinal tissue or fluid; (2) evidence of mediastinitis seen during an operation; (3) one of the following conditions: chest pain, sternal instability, or fever (>38 · C), *in combination with* either purulent discharge from the mediastinum or an organism isolated from blood culture or culture of mediastinal drainage.

**Pneumonia:** Pneumonia diagnosed by one of the following: Positive cultures of sputum, blood, pleural fluid, emphysema fluid, transtracheal fluid or transthoracic fluid; consistent with the diagnosis and clinical findings of pneumonia. Should include chest x-ray diagnostic of pulmonary infiltrates.




**Sepsis:** Culture-proven blood infection manifested by severe systemic symptoms (e.g. fever, hyperventilation, tachycardia, confusion).

**Septic Shock:** Sepsis with hypotension despite adequate fluid resuscitation. In addition, two or more of the following must be present:

- tachycardia
- temperature < 36° or > 38°C
- hyperventilation
- WBC < 4000 or > 12000

**Urinary Tract Infection:** Positive urine cultures requiring antibiotic therapy.

**Viral Illness:** Diseases caused by a virus, including Bronchitis, Sinusitis, Cellulitis, and Upper Respiratory Infection.

# INJURY, POISONING AND PROCEDURAL COMPLICATIONS

**Atrial Tear**: Any evidence of a tear or damage to the two upper chambers of heart/atrium

**Cardiac Valve Injury:** Damage to any cardiac valve resulting from the index hybrid surgical procedure.

Coronary Artery Injury: Damage to the artery caused during surgery requiring repair.

**Dissections**: Presence of angiographically evident intimal disruption (e.g., linear luminal density or luminal staining or linear intraluminal filling defect) which requires treatment.

**Ventricular Perforation or Rupture:** Any evidence of puncture/dissection/perforation or damage to the ventricle.

**Pseudoaneurysm**: Compartmentalized blood contiguous with arterial lumen documented by ultrasound or visualized at repair.

# Skin Burns:

- **Second degree burns** manifest as erythema with superficial blistering of the skin. Level of pain is dependent upon the level of nerve involvement.
- **Third-degree burns:** occur when the epidermis is lost with damage to the subcutaneous tissue. This burn may exhibit charring and extreme damage of the epidermis, and sometimes hard eschar will be present.

Wound dehiscence/delayed wound healing: not associated with infection.




# **METABOLISM DISORDERS**

**Hyperglycemia:** The use of insulin in the post op period does not constitute hyperglycemia if during the same hospitalization. An Elevated blood sugar ≥ 250 in the post-operative constitutes hyperglycemia.

**Hypoglycemia**: Low blood glucose or low blood sugar, occurs when blood glucose drops below normal levels (50mg/dL).

# **NERVOUS SYSTEM DISORDERS**

**Headache:** a term used to describe aching or pain that occurs in one or more areas of the head, face, mouth, or neck. Headache can be chronic, recurrent, or occasional.

**Recurrent Laryngeal Nerve Injury**: Symptomatic hoarseness with documented laryngoscopy showing paralyzed or impaired laryngeal cord movement, beyond 30 days post procedure.

**Phrenic Nerve Paralysis:** Phrenic nerve paralysis is defined as absent phrenic nerve function as assessed by a sniff test. A phrenic nerve paralysis is considered to be permanent when it is documented to be present at 12 months or longer following ablation.

**Seizures**: sudden, uncontrolled muscle spasms with or without loss of consciousness resulting from brain electrical activity

**Stroke:** Rapid onset of a focal or global neurological deficit with at least one of the following: change in level of consciousness, hemiplegia, hemiparesis, numbness or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopia, amaurosis fugax, or other neurological signs or symptoms consistent with stroke. Duration of neurological deficit lasting ≥ 24 hours, or lasting <24 hours if therapeutic intervention(s) were performed (i.e. thrombolytic therapy or intracranial angioplasty; or available neuro imaging documents a new hemorrhage or infarct or the neurological deficit results in death. Confirmation of the diagnosis by at least one of the following; neurology or neurosurgical specialist, neuro imaging study showing tissue injury or lumbar puncture demonstrating intracranial hemorrhage.

Stroke diagnosis will be performed preferably with positive neuroimaging study. The stroke will be assessed as Minor or Major based on the following:

- Minor—Modified Rankin (mRS) score <2 at 30 and 90 days</li>
- Major—Modified Rankin (mRS) score >2 at 30 and 90 days

May be further categorized as:

• Ischemic Stroke: Neurologic deficit attributed to thromboembolic event.




 Hemorrhagic Stroke: Neurologic deficit meeting the study definition for Stroke that is attributed to bleeding into brain tissue, epidural, subdural, or subarachnoid space; or a combination of these sites

**Systemic Embolism:** The obstruction of blood flow in a vessel by an embolus (which may include a thrombus or an air bubble), in the pulmonary or peripheral arterial circulation. Diagnosis must be confirmed on imaging study, and interventional treatment performed to address condition. Does not include neurologic events (See Stroke definition).

**Transient Ischemic Attack (TIA):** Neurological deficit lasting less than 24 hours and, if an imaging study is performed, shows no evidence of infarction.

Vagal Nerve Injury: see esophageal dyskinesia and gastroparesis

**Vasovagal Reaction:** Reflex stimulation of the vagus nerve causing slowing of the heartbeat, decreased blood pressure, etc. and requires treatment consisting of any of the following: (a) > 1 liter of IV fluids; (b) postural changes; (c) pacing intervention; or (d) administration of atropine.

### **PSYCHIATRIC DISORDERS**

**Anxiety:** A psychiatric disorder causing feelings of mental discomfort, for example, panic disorder, post-traumatic stress disorder or depression.

# RESPIRATORY/PULMONARY

**Acute respiratory distress syndrome (ARDS):** A failure of the respiratory system characterized by fluid accumulation within the lung that causes the lung to stiffen. This condition must be confirmed by radiological evidence, or lung biopsy, or the need for prolonged positive pressure ventilation.

**Atelectasis:** (post-surgical) is a collapse of lung tissue affecting part or all of one lung; the alveoli are deflated. This is an AE when treatment other than Chest PT is required or it prolongs hospitalization.

**Diaphragmatic paralysis:** may be unilateral or bilateral. Usually caused by injury to the phrenic nerve as a result of trauma to the thoracic cage. Findings include decreased air flow, dullness to percussion, and absence of diaphragmatic excursion on the ipsilateral side. Diagnosis may be made with fluoroscopy in which a quick "sniff" (i.e. subject inspiration) results in observation of paradoxical elevation of the ipsilateral diaphragm. Often causes shortness of breath on activity.

**Hemoptysis:** A cough that produces bloody sputum.




**Pleural Effusion**: Accumulation of fluid in the pleural space evidenced by x-ray, echocardiography, CT Scan or other appropriate diagnostic technique and which requires drainage.

**Pneumothorax:** Air in the thoracic cavity associated with partial collapse of a lung with chest tube drainage required.

**Pulmonary Edema:** Pulmonary edema is present if there is fluid accumulation in the lungs caused by backpressure in the lung veins. This condition must be confirmed by radiological evidence or lung water measurements.

**Pulmonary Embolism**: Pulmonary embolism diagnosed by study such as V/Q scan or angiogram or spiral CT or clinical symptoms consistent with PE in the absence of these studies that result in treatment.

**Pulmonary Hypertension**: Subject has mean pulmonary artery pressure that is greater than 25 mmHg at rest and/or greater than 30 mmHg during exercise as measured by right heart catheterization.

**Pulmonary vein stenosis:** Defined as 70% diameter stenosis of one pulmonary vein or 50% diameter stenosis of more than one vessel. PV stenosis is manifest as dyspnea at rest, may be associated with hemoptysis and must be confirmed by imaging studies of the pulmonary veins (using CT or MRI).

**Respiratory failure:** Need for mechanical ventilation beyond 48 hours of completion of surgical procedure(s), or the need for re-intubation and ventilator support occurring at any time within 30 days of the surgical procedure, outside the setting of an additional operation.

**Respiratory insufficiency**: Deterioration of subject's respiratory efforts that require supportive or medical treatment.

#### **VASCULAR DEFINITIONS**

Atrial Embolism: Angiographic evidence of embolic occlusion in any arterial distribution.

**Arterial Occlusion/Thrombosis at Access Site**: Angiographic or ultrasonographic evidence of occlusion at the access site,

**Arteriovenous Fistula**: A traumatic communication between an artery and vein documented by ultrasound or angiography




**Deep Vein Thrombosis (DVT)**: Angiographic or ultrasonographic evidence of thromboembolic occlusion in the lower extremities.

**Embolism (including air emboli and thromboemboli)**: The blockage of an artery by an embolus, which can include a thrombus or an air bubble.

**Hematoma**: Development of a collection of blood > 5 cm under the skin requiring compression or additional treatment to resolve.

**Major Bleeding:** The following will constitute major bleeding events:

- Fatal bleeding OR
- Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome OR
- Bleeding causing hypovolemic shock or severe hypotension requiring surgery OR
- Overt source of bleeding with drop in hemoglobin ≥5 g/dL or whole blood or packed red blood cells (RBCs) transfusion ≥4 units

**Hypertension:** Systolic BP > 140 mmHg, or diastolic > 90 mmHg, or requiring specific medical therapy.

**Hypotension:** Any prolonged systolic blood pressure < 80 mmHg associated with symptoms and requiring intravenous vasopressor medications.

**Limb Ischemia**: Limb ischemia is manifested by pain in an extremity at rest, associated with non-healing wounds and gangrene. Limb ischemia should be confirmed by diagnostic imaging studies.

**Peripheral Ischemia**: Deficient supply of blood to the blood vessels outside the heart and brain that is due to obstruction of the inflow of arterial blood.

**Thromboembolism**: Formation of a thrombus (*masses composed of insoluble fibrin, deposited platelets, accumulating WBCs, and entrapped RBCs*) that obstructs vascular blood flow locally and detaches and embolizes to occlude blood flow downstream. Diagnostic confirmation should be made with angiography or ultrasound.

**Thrombophlebitis:** Inflammation of a vein with formation of a thrombus.

**Thrombus**: Blood clot that obstructs a blood vessel.




# APPENDIX IV: FORSEEABLE ADVERSE EVENTS

Adverse Events that may be anticipated in this clinical study are believed to be consistent with those associated with other invasive surgical and cardiac procedures.

Complications that may have occurred at any time during the procedure, post procedure or that are possible during the follow-up period with the AtriCure AtriClip LAA Exclusion System include, but are not limited to the following:

- Air embolism
- Allergic reaction to implant materials
- Anesthesia risks
- Aneurysm
- Angina
- Arrhythmia needing medical treatment (new onset)
- Arterial or venous dissection and/or perforation
- Arterial rupture
- Arterial spasm
- Arteriovenous fistula
- Atelectasis (major lung tissue collapse with significant symptoms such as cyanosis, extreme shortness of breath, dyspnea, and/or stabbing pain on the affected side)
- Atrial rupture
- AV block requiring permanent pacemaker (new onset)
- Bleeding requiring intervention to repair or which requires > 2 units of blood products
- Blood vessel damage
- Cardiac perforation
- Cardiac tamponade (if either open chest or catheter drainage is required)
- Coronary artery injury
- Cardiac valve injury
- Cerebrovascular accident (CVA)/stroke (ischemic or hemorrhagic)
- Circumflex artery impingement
- Conduction disturbances (SA/AV node)
- Congestive heart failure (new onset or exacerbation)
- Death
- Diaphragmatic paralysis (unilateral or bilateral)
- Drug Reaction (significant reaction to any study related medications requiring treatment, including allergic reaction and anaphylactic shock)
- Emergency during the operation requiring change in the planned surgical access
- Endocarditis (bacterial)




- Pain and discomfort
- Extension of cardiopulmonary/extracorporeal bypass
- Esophageal rupture
- Extravasation of contrast media
- Fever
- Gastro-intestinal bleed
- · Gastric motility disorders
- Hematoma
- Hematuria
- Hemothorax
- Hypertension
- Hypotension
- latrogenic lung injury (e.g., chest tube placement)
- Infection requiring treatment
- Injury to the heart, a blood vessel, or other part of the body due to the investigational device, possibly requiring intervention
- Ischemia
- Myocardial infarction (MI)
- Nerve Injury (phrenic, laryngeal, thoracic, etc.)
- Pericarditis
- Persistent chest pain (post discharge surgical incision pain, not angina)
- Pericardial effusion
- Pleural effusion
- Pneumothorax (requiring intervention)
- Postoperative embolic complications
- Pseudoaneurysm
- Pulmonary edema
- Pulmonary embolism
- Renal insufficiency or failure
- Respiratory distress or failure (breathing problems)
- Sepsis
- Sinus Node Dysfunction (new onset)
- Thrombus and/or thromboembolism (including a deep vein thrombosis)
- Transient ischemic attack (TIA)
- Tracheal esophageal trauma
- Unanticipated device effects
- There may also be other risks that are unforeseen at this time.




# **APPENDIX V: INFORMED CONSENT FORM**

A copy of the Sponsor Informed Consent Form Template can be obtained upon request from the Sponsor Clinical Project Manager for the clinical investigation and will be provided to study sites for IRB/EC approval.






# **APPENDIX VI: SITE CONTACT INFORMATION**

A copy of contact information for each participating site can be obtained upon request from the Sponsor Clinical Project Manager for the clinical investigation.






# **APPENDIX VII: REVISION HISTORY**

| Amendment<br>Number | Version /<br>Revision | Details |
|---|---|---|
| Not Applicable | RCS-036<br>rev. A | Initial Release per DCN-2021-0640. |
| Not Applicable | CP-2021-<br>03 rev. B | See redlines on DCN-2021-0738 for all changes. Changes include: • Protocol number changed from RCS-036 to CP-2021-03 to match CP number in other literature. • Protocol revised due to a need to change performance goals to better reflect contemporary literature for LAA closure rates. |

